**Protocol Number: AVXS-101-CL-302** 

Official Title: Phase 3, Open-Label, Single-Arm, Single-Dose Gene
Replacement Therapy Clinical Trial for Patients with Spinal
Muscular Atrophy Type 1 with One or Two SMN2 Copies
Delivering AVXS-101 by Intravenous Infusion

NCT Number: NCT03461289

Document Date: 25-Jun-2020

# SIGNATURE PAGE TITLE CL-302 Clinical Protocol ID: PRO-747

| User | Role | Job Title | Version | Decision | Date Signed |
|---|---|---|---|---|---|
| | Final Approvers | Senior Director, U.S. Regulatory<br>Affairs | 7.0 | Approve | 03 Jul 2020 06:41 PM<br>CEST |
| | Final Approvers | Executive Medical Director | 7.0 | Approve | 03 Jul 2020 08:03 PM<br>CEST |
| | Final Approvers | Associate Director, Therapeutic<br>Lead | 7.0 | Approve | 03 Jul 2020 05:27 PM<br>CEST |
| | Final Approvers | Sr Dir. Clinical Development (EMEA) | 7.0 | Approve | 03 Jul 2020 06:36 PM<br>CEST |
| | Final Approvers | Vice President | 7.0 | Approve | 03 Jul 2020 06:50 PM<br>CEST |
| | Final Approvers | Senior Director, Biostatistics | 7.0 | Approve | 03 Jul 2020 06:48 PM<br>CEST |

This is a copy generated on 22 Sep 2020 08:42 PM CEST. Please refer to ACE for most recent effective version.



# AVXS-101 AVXS-101-CL-302

**IND Number:** 15699

**EudraCT Numbers:** 2017-000266-29

**Protocol Title:** Phase 3, Open-Label, Single-Arm, Single-Dose Gene

Replacement Therapy Clinical Trial for Patients with Spinal Muscular Atrophy Type 1 with One or Two *SMN2* Copies

Delivering AVXS-101 by Intravenous Infusion

**Indication Studied:** Spinal Muscular Atrophy Type 1

**Sponsor Address:** AveXis, Inc.

2275 Half Day Road, Suite 200

Bannockburn, IL 60015

**Protocol Version/Date:** 7.0/Amendment 6/25 Jun 2020

The trial will be completed according to the guidelines of Good Clinical Practice. Compliance with this standard provides public assurance that the rights, safety, and well-being of trial subjects are protected, consistent with the principles that have their origin in the Declaration of Helsinki.

# **Confidentiality Statement**

The information in this document contains trade and commercial information that is privileged or confidential and may not be disclosed unless such disclosure is required by federal or state law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may

not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you which is indicated as privileged or confidential.

Investigational Product: AVXS-101 Protocol Version 7.0/Amendment 6/25 Jun 2020

#### 1. ADMINISTRATIVE INFORMATION

# 1.1. Approval

## **Representatives from AveXis:**

This trial will be conducted with the highest respect for the individual participants in accordance with the requirements of this clinical trial protocol and also in accordance with the following:

- The ethical principles that have their origin in the Declaration of Helsinki
- International Council for Harmonisation, Integrated Addendum to ICH E6 (R1): Guideline for Good Clinical Practice E6 (R2)
- All applicable laws and regulations, including, without limitation, data privacy laws and regulations

SIGNATURES (may be applied electronically and will therefore be maintained in the electronic system):

| Vice President, Clinical Development & Analytics<br>AveXis, Inc. | Date (ddMmmyyyy) |
|---|---|
| Senior Director, Clinical Development<br>AveXis, Inc. | Date (ddMmmyyyy) |
| Senior Director, Regulatory Affairs<br>AveXis, Inc. | Date (ddMmmyyyy) |
| Associate Director, Therapeutic Lead<br>AveXis, Inc. | Date (ddMmmyyyy) |
| Senior Director, Biostatistics<br>AveXis, Inc. | Date (ddMmmyyyy) |
| Vice President & Head, Global Patient Safety<br>AveXis, Inc. | Date (ddMmmyyyy) |

Investigational Product: AVXS-101

Protocol Version 7.0/Amendment 6/25 Jun 2020

# 1.2. Investigator's Agreement

I have received and read the Investigator's Brochure for AVXS-101. I have read the AVXS-101-CL-302 protocol and agree to conduct the trial in accordance with the relevant current protocol.

I agree to maintain the confidentiality of all information received or developed in connection with this protocol. I agree to personally conduct or supervise the investigation(s). I also agree to promptly report to the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) all changes in the research activity and all unanticipated problems involving risks to human subjects or others. Additionally, I will not make any changes in the research without IRB/IEC approval, except where necessary to eliminate apparent immediate hazards to human subjects. I agree to protect the safety, rights, privacy, and well-being of trial participants. I agree to comply with:

- The ethical principles that have their origin in the Declaration of Helsinki
- International Council for Harmonisation, Integrated Addendum to ICH E6 (R1): Guideline for Good Clinical Practice E6 (R2)
- All applicable laws and regulations, including, without limitation, data privacy laws and regulations including but not limited to Clinical Trials Directive 2001/20/EC and Regulation (European Union) No 536/2014 of the European Parliament and of the Council of 16 April 2014 on clinical trials of medicinal products for human use
- Terms outlined in the trial site agreement
- Responsibilities of the Investigator (per regulatory guidelines and applicable regulations)

I further authorize that my personal information may be processed and transferred in accordance with the uses contemplated in this protocol.

# **Confidentiality Statement**

The confidential information in this document is provided to you as a Principal Investigator or Consultant for review by you, your staff, and the applicable Institutional Review Board/Independent Ethics Committee. Your acceptance of this document constitutes agreement that you will not disclose the information contained herein to others without written authorization from the Sponsor.

| Printed Name of Principal Investigator |
|----------------------------------------|
| Timos Timos par mi verigaren |
| Signature of Principal Investigator |
| Signature of Finicipal Investigator |

PRO-747 Version7.0 Generated 22 Sep 2020 08:42 PM CEST | Effective Date: 03 Jul 2020 08:04 PM CEST

AveXis, Inc.

AVXS-101-CL-302

Investigational Product: AVXS-101


Date (ddMmmyyyy)

Investigational Product: AVXS-101


# 1.3. Key Contact Information

| Role in Study | Contact Information |
|------------------------------------|---------------------------------------|
| Responsible Physician | Senior Director, Clinical Development |
| Serious Adverse Event<br>Reporting | E-mail: Fax: |

Additional study contact information is provided in the Study Contact List.


#### 2. SYNOPSIS

Name of Sponsor/Company: AveXis, Inc.

Name of Investigational Product: AVXS-101

Name of Active Ingredient: Survival Motor Neuron Gene by Self-Complementary Adeno-Associated

Virus Serotype 9 (AAV9)

**Title of Trial:** Phase 3, Open-Label, Single-Arm, Single-Dose Gene Replacement Therapy Clinical Trial for Patients with Spinal Muscular Atrophy Type 1 with One or Two *SMN2* Copies Delivering AVXS-101 by Intravenous Infusion

**Estimated number of Trial Center(s) and Countries or Regions:** 12–16 European Investigative Sites located in the following countries: Belgium, France, Germany, Italy, Netherlands, Spain, United Kingdom, Sweden

Phase of Development: 3

Investigators: Multicenter Trial - Investigator Information on File at AveXis

#### **Studied Period (years):**

Estimated date first patient enrolled: Q2 2018 Estimated date last patient completed: Q3 2020

#### **Objectives: Primary**

 Determine efficacy by demonstrating achievement of developmental milestone of sitting without support for at least 10 seconds up to 18 months of age as defined by WHO Motor Developmental Milestone.

#### **Secondary**

Determine efficacy based on survival at 14 months of age. Survival is defined by the avoidance of combined endpoint of either (a) death or (b) permanent ventilation which is defined by tracheostomy or by the requirement of ≥ 16 hours of respiratory assistance per day (via non-invasive ventilatory support) for ≥ 14 consecutive days in the absence of an acute reversible illness, excluding perioperative ventilation. Permanent ventilation, so defined, is considered a surrogate for death.

#### **Exploratory**

 Determine efficacy by demonstrating achievement of developmental milestone of ability to hold head erect without support as defined by Bayley Scales of Infant and Toddler Development© Version 3 (BSIDv03) Gross Motor Subtest Item #4.


- Determine efficacy by demonstrating achievement of developmental milestone of ability to roll over as defined by BSIDv03 Gross Motor Subtest Item #20.
- Determine the efficacy by demonstrating achievement of developmental milestone of functional independent sitting for at least 30 seconds as defined by BSIDv03 Gross Motor Subtest Item #26.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand with assistance for at least 2 seconds as defined by BSIDv03 Gross Motor Subtest Item #33.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to crawl forwards on hands and knees for a distance of at least 5 feet as defined by BSIDv03 Gross Motor Subtest Item #34.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to pull to standing as defined by BSIDv03 Gross Motor Subtest Item #35.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk with assistance as defined by BSIDv03 Gross Motor Subtest Item #37.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand alone for at least 3 seconds as defined by BSIDv03 Gross Motor Subtest Item #40.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk at least 3 steps without support as defined by BSIDv03 Gross Motor Subtest Item #42.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to crawlas defined by WHO Motor Developmental Milestones.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand with assistance as defined by WHO Motor Developmental Milestones.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand alone as defined by WHO Motor Developmental Milestones.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk with assistance as defined by WHO Motor Developmental Milestones.
- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk alone as defined by WHO Motor Developmental Milestones.
- Determine efficacy by demonstrating improvement of motor function as determined by improvement in the fine and gross motor domain components of the Bayley Scales of Infant and Toddler Development© (Version 3).
- Determine efficacy by demonstrating improvement of gross motor function as determined by improvement in Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) score.


- Determine the effect of AVXS-101 on the ability to remain independent of ventilator support, defined as requiring no daily ventilator support/usage at 18 months of age.
- Determine effect on the ability to thrive defined as achieving all of the following:
  - Does not receive nutrition through mechanical support (i.e., feeding tube)
  - Ability to tolerate thin liquids as demonstrated through a formal swallowing test
  - Maintains weight (> third percentile for age and gender).

#### Safety

Evaluate the safety of AVXS-101 in patients with SMA Type 1.

#### Methodology:

Phase 3, open-label, single-arm, single-dose, trial of AVXS-101 (gene replacement therapy) in patients with spinal muscular atrophy (SMA) Type 1 who meet enrollment criteria and are genetically defined by a biallelic pathogenic mutation of the survival motor neuron 1 gene (SMN1) with 1 or 2 copies of survival motor neuron 2 gene (SMN2). Thirty patients < 6 months (< 180 days) of age <u>at the time</u> of gene replacement therapy (Day 1) are planned to be enrolled.

The trial includes a screening period, a gene replacement therapy period, and a follow-up period. During the screening period (Days –30 to –2), patients whose parent(s)/legal guardian(s) provide informed consent will complete screening procedures to determine eligibility for trial enrollment. Patients who meet the entry criteria will enter the in-patient gene replacement therapy period (Day –1 to Day 3). On Day –1, patients will be admitted to the hospital for pre-treatment baseline procedures. On Day 1, patients will receive a 1-time intravenous (IV) infusion of AVXS-101 and will undergo inpatient safety monitoring over the next 48 hours. Patients may be discharged 48 hours after the infusion, based on Investigator judgment. During the outpatient follow-up period (Days 4 to End of Trial at 18 months of age), patients will return at regularly scheduled intervals for efficacy and safety assessments until the End of Trial when the patient reaches 18 months of age. After the End of Trial visit, patients will be invited to participate in a long-term follow up study conducted under a separate protocol. Patients who discontinue the trial prematurely will also be invited to participate in the long-term follow up study.

All post-treatment visits will be relative to the date on which gene replacement therapy is administered until the patient is 14 months of age, after which all visits will be relative to the patient's date of birth.

In an attempt to dampen the host immune response to the adeno-associated virus (AAV) derived therapy, all patients will receive prophylactic prednisolone at approximately 2 mg/kg/day (or an equivalent dose of another glucocorticoid if prednisolone is unavailable or in the opinion of the investigator prednisolone is not tolerated [39]) on Day -1, Day 1, and Day 2, and then 1 mg/kg/day starting on Day 3 and until at least 30 days post-AVXS-101 infusion. After 30 days post-AVXS-101 infusion, the dose of prednisolone can be tapered for patients whose gamma glutamyl transferase (GGT), alanine aminotransferase (ALT) values, and aspartate aminotransferase (AST) values are below

Investigational Product: AVXS-101


the threshold of 2  $\times$  Upper Limit Normal (ULN) in accordance with the following treatment guideline: taper from 1 mg/kg/Day to 0.5 mg/kg/Day during Weeks 5 and 6 post-AVXS-101 infusion, then taper to 0.25 mg/kg/Day during Weeks 7 and 8, and then discontinue prednisolone at Week 9. If the AST or ALT values are  $> 2 \times$  ULN, the dose of prednisolone will be maintained until the AST and ALT values decrease below threshold. Variance from these recommendations will be at the discretion of the Investigator based on potential safety issues for each patient. If another glucocorticoid is used in place of prednisolone by the Investigator, similar considerations should be taken into account after 30 days and tapered as appropriate and at the discretion of the Investigator.

Efficacy will be assessed by achievement of the key developmental milestone of sitting without support for at least 10 seconds based on World Health Organization [WHO] Child Growth Standards at any point up to and including the 18 months of age trial visit, and survival at 14 months of age.

Safety will be assessed through monitoring adverse events (AEs), concomitant medication usage, physical examinations, vital sign assessments, cardiac assessments, and laboratory evaluations. A Data Safety Monitoring Board (DSMB)/Data Monitoring Committee (DMC) will review safety data on a quarterly basis and will also convene within approximately 48 hours should any patient experience an unanticipated CTCAE Grade 3, or higher AE/toxicity that is possibly, probably, or definitely related to gene replacement therapy, and is associated with clinical symptoms and/or requires medical treatment. This includes any patient death, important clinical laboratory finding, or any complication attributed to administration of gene replacement therapy. In such instances, the DSMB/DMC will review the safety information and provide its recommendation. Based upon the DSMB/DMC's review, the DSMB/DMC can recommend continuing enrollment, halting enrollment, or early termination of the trial for safety reasons.

**Number of Patients (planned):** Thirty patients are planned to enroll. Babies who are in screening and meet eligibility criteria for the study when the enrollment target is met may be enrolled upon approval of the sponsor.

#### Diagnosis and Main Criteria for Inclusion: Inclusion Criteria:

- 1. Patients with SMA Type 1 as determined by the diagnosis of SMA based on gene mutation analysis with biallelic *SMN1* mutations (deletion or point mutations) and 1 or 2 copies of *SMN2* [inclusive of the known *SMN2* gene modifier mutation (c.859G>C)]
- 2. Patients must be < 6 months (< 180 days) of age at the time of AVXS-101 infusion.
- 3. Patients must have a swallowing evaluation test performed prior to administration of gene replacement therapy.
- 4. Up-to-date on childhood vaccinations that include palivizumab prophylaxis (also known as Synagis) to prevent respiratory syncytial virus (RSV) infections are also recommended.
- 5. Parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with trial procedures and visit schedule.

#### **Exclusion Criteria:**


- 1. Previous, planned or expected scoliosis repair surgery/procedure prior to 18 months of age.
- 2. Use of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry < 95% saturation at screening
  - a. Pulse oximetry saturation must not decrease ≥ 4 percentage points between screening and dosing with confirmatory oximetry reading
  - b. Patients may be put on non-invasive ventilatory support for < 12 hours per day at the discretion of their physician or trial staff.
- 3. Use or requirement of non-invasive ventilatory support for ≥12 hours daily in the 2 weeks prior to dosing.
- 4. Patient with signs of aspiration based on a swallowing test or whose weight-for-age falls below the 3<sup>rd</sup> percentile based on World Health Organization (WHO) Child Growth Standards and is unwilling to use an alternative method to oral feeding.
- 5. Active viral infection (includes human immunodeficiency virus [HIV] or positive serology for hepatitis B or C or known Zika virus infection).
- 6. Serious non-respiratory tract illness requiring systemic treatment and/or hospitalization within 2 weeks prior to screening.
- 7. Upper or lower respiratory infection requiring medical attention, medical intervention, or increase in supportive care of any manner within 4 weeks prior to screening.
- 8. Severe non-pulmonary/respiratory tract infection (e.g., pyelonephritis, or meningitis) within 4 weeks before administration of gene replacement therapy or concomitant illness that, in the opinion of the Principal Investigator, creates unnecessary risks for gene replacement such as:
  - a. Major renal or hepatic impairment
  - b. Known seizure disorder
  - c. Diabetes mellitus
  - d. Idiopathic hypocalciuria
  - e. Symptomatic cardiomyopathy.
- 9. Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients.
- 10. Concomitant use of any of the following: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, or immunosuppressive therapy within 3 months prior to gene replacement therapy (e.g., corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, IV immunoglobulin, rituximab).
- 11. Anti-AAV9 antibody titer > 1:50 as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay. Should a potential patient demonstrate Anti-AAV9 antibody titer > 1:50,

Investigational Product: AVXS-101


he or she may receive retesting within 30 days of the screening period and will be eligible to participate if the Anti-AAV9 antibody titer upon retesting is  $\leq 1:50$ .

- 12. Clinically significant abnormal laboratory values (gamma-glutamyl transpeptidase [GGT], alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin > 2 × the upper limit of normal (ULN), creatinine ≥ 1.0 mg/dL, hemoglobin [Hgb] < 8 or > 18 g/dL; white blood cell [WBC] > 20,000 per cmm) prior to gene replacement therapy. Patients with an elevated bilirubin level that is unequivocally the result of neonatal jaundice shall not be excluded.
- 13. Participation in recent SMA treatment clinical trial (with the exception of observational Cohort studies or non-interventional studies) or receipt of an investigational or commercial compound, product or therapy administered with the intent to treat SMA (e.g., nusinersen, valproic acid,) at any time prior to screening for this trial. Oral  $\beta$ -agonists must be discontinued at least 30 days before gene therapy dosing. Inhaled albuterol specifically prescribed for the purposes of respiratory (bronchodilator) management is acceptable and not a contraindication at any time prior to screening for this trial.
- 14. Expectation of major surgical procedures during the trial assessment period (e.g., spinal surgery or tracheostomy).
- 15. Parent(s)/legal guardian(s) unable or unwilling to comply with trial procedures or inability to travel for repeat visits.
- 16. Parent(s)/legal guardian(s) unwilling to keep trial results/observations confidential or to refrain from posting confidential trial results/observations on social media sites.
- 17. Parent(s)/legal guardian(s) refuses to sign consent form.
- 18. Patient < 35 weeks gestational age at time of birth.

#### **Investigational Product, Dosage and Mode of Administration:**

Patients will receive a 1-time dose of AVXS-101 at  $1.1 \times 10^{14}$  vg/kg, a dose determined to be equivalent to the dose received by the Cohort 2 patients in the Phase 1 study (AVXS-101-CL-101) by direct testing using improved analytical methods.

#### **Duration of Treatment:**

AVXS-101 will be administered as a 1-time IV infusion over 60 minutes, dependent upon volume.

Reference Therapy, Dosage and Mode of Administration: Not Applicable

#### **Endpoint: Efficacy:**

#### **Primary**

Proportion of symptomatic SMA Type 1 patients who are homozygous negative for SMN1 exon
 7 and have 2 copies of SMN2 without the SMN2 genetic modifier that achieve the ability to sit

Investigational Product: AVXS-101


without support for at least 10 seconds up to and including the 18 months of age trial visit. Sitting without support is defined by the World Health Organization Multicentre Growth Reference Trial (WHO MGRS), confirmed by video recording, as a patient who sits up straight with head erect for at least 10 seconds; child does not use arms or hands to balance body or support position.

#### Secondary

• Survival at 14 months of age amongst symptomatic SMA Type 1 patients who are homozygous negative for SMN1 exon 7 and have 2 copies of SMN2 without the SMN2 genetic modifier. Survival is defined by the avoidance of the combined endpoint of either (a) death or (b) permanent ventilation, which is defined by tracheostomy or by the requirement of ≥ 16 hours of respiratory assistance per day (via non-invasive ventilatory support) for ≥ 14 consecutive days in the absence of an acute reversible illness, excluding perioperative ventilation. Permanent ventilation, so defined, is considered a surrogate for death.

#### **Exploratory**

- Proportion of patients that achieve the ability to hold head erect without support as defined by BSIDv03 Gross Motor Subtest Item #4.
- Proportion of patients that achieve the ability to roll over as defined by BSIDv03 Gross Motor Subtest Item #20.
- Proportion of patients that achieve functional independent sitting for at least 30 seconds as defined by BSIDv03 Gross Motor Subtest Item #26.
- Proportion of patients that achieve the ability to stand with assistance for at least 2 seconds as defined by BSIDv03 Gross Motor Subtest Item #33.
- Proportion of patients that achieve the ability to crawl forwards on hands and knees for a distance of at least 5 feet as defined by BSIDv03 Gross Motor Subtest Item #34.
- Proportion of patients that achieve the ability to pull to standing as defined by BSIDv03 Gross Motor Subtest Item #35.
- Proportion of patients that achieve the ability to walk with assistance as defined by BSIDv03 Gross Motor Subtest Item #37.
- Proportion of patients that achieve the ability to stand alone for at least 3 seconds as defined by BSIDv03 Gross Motor Subtest Item #40.
- Proportion of patients that achieve the ability to walk at least 3 steps without support as defined by BSIDv03 Gross Motor Subtest Item #42.
- Proportion of patients that achieve the ability to crawl as defined by WHO Motor Developmental Milestones.
- Proportion of patients that achieve the ability to stand with assistance as defined by WHO Motor Developmental Milestones.


- Proportion of patients that achieve the ability to stand alone as defined by WHO Motor Developmental Milestones.
- Proportion of patients that achieve the ability to walk with assistance as defined by WHO Motor Developmental Milestones.
- Proportion of patients that achieve the ability to walk alone as defined by WHO Motor Developmental Milestones.
- Improvement of raw score from baseline to the maximum using Bayley Scales of Infant and Toddler Development (Version 3), Fine and Gross Motor Function Subtests.
- Maximum change from baseline of CHOP INTEND score.
- Proportion of patients achieving CHOP INTEND score ≥ 40.
- Proportion of patients achieving CHOP INTEND score ≥ 50.
- Proportion of patients achieving CHOP INTEND score ≥ 58.
- Proportion of patients with the ability to remain independent of ventilator support, defined as requiring no daily ventilator support/usage at 18 months of age.
- Proportion of patients maintaining the ability to swallow and to maintain weight
   (> 3<sup>rd</sup> percentile based on WHO Child Growth Standards for age and gender) without need of
   gastrostomy or other mechanical or non-oral nutritional support.
- Age at which (WHO MGRS) sitting without support (10 seconds) is first achieved.

#### **Endpoint Safety:**

Assessment of the safety and tolerability of AVXS-101 treatment includes evaluation of AEs, laboratory data, vital signs, and concomitant medications.

#### **Statistical Methods:**

This is a pivotal Phase 3 trial assessing the efficacy and safety of AVXS-101. Details of all analysis will be contained within the Statistical Analysis Plan.

The primary and secondary efficacy analyses will be performed amongst symptomatic patients with biallelic *SMN1* deletions and 2 copies of *SMN2* without the genetic modifier (c.859G>C). While the study will enroll a small number of additional patients, the above will comprise the population for evaluation of the primary and secondary endpoints and will be referred to as the ITT population hereafter.

Based upon widely cited natural history of the disease (Pediatric Neuromuscular Clinical Research Network [PNCR]), it is expected that no patients in this population would be expected

Investigational Product: AVXS-101


to attain the ability to sit without support or attain other developmental milestones (rolling over, standing, walking) assessed as part of the trial.

Assuming that the true response rate for the primary endpoint is actually zero (or as low as 0.1%) in the population of interest of the historical control, the primary efficacy endpoint hypothesis is whether AVXS-101 treated patients achieve a response rate greater than 0.1%.

Based upon preliminary results from the completed Phase 1 clinical trial AVXS-101-CL-101, at least 50% of treated patients in the defined ITT population are expected to achieve the primary efficacy endpoint of sitting without support for at least 10 seconds at any post-procedure visit up to and including 18 months of age. With this assumption for the true response rate of AVXS-101 being in the range of 20%–50%, a sample size of 25 patients would provide power of greater than 95% to detect a significant difference from 0.1% with  $\alpha$  = 0.025 using a 1-sided exact test for a binomial proportion.

The secondary efficacy endpoint of survival at 14 months of age will be comparing the results observed in the ITT population with the results from the age and gender-matched control patients selected from existing natural history data sets (PNCR). It is anticipated that 75% of patients in the PNCR population would not survive beyond 13.6 months of age, and that these control patients will represent a 25% survival rate based upon the natural history of the disease. Preliminary results from the completed Phase I clinical study, AVXS-101-CL-101, suggest that at least 80% of patients in the ITT population are expected to survive, as defined, through 14 months of age. These assumptions suggest that a sample size of at least 25 patients would provide at least 95% power to detect a significant difference from the historical control with  $\alpha$  = 0.05 using a 2-sided Fisher's Exact test.

Investigational Product: AVXS-101

#### Protocol Version 7.0/Amendment 6/25 Jun 2020

# 3. TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES

# **TABLE OF CONTENTS**

| 1. | ADMINISTRATIVE INFORMATION | 3 |
|------|--------------------------------------------------------|----|
| 1.1. | Approval | 3 |
| 1.2. | Investigator's Agreement | |
| 1.3. | Key Contact Information | 6 |
| 2. | SYNOPSIS | |
| 3. | TABLE OF CONTENTS, LIST OF TABLES, AND LIST OF FIGURES | 16 |
| 4. | LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS | 21 |
| 5. | INTRODUCTION | 24 |
| 5.1. | Background | 24 |
| 5.2. | Rationale for Gene Transfer to SMA Type 1 Patients | 25 |
| 5.3. | Nonclinical Studies | 27 |
| 5.4. | Clinical Studies | 31 |
| 5.5. | Risks | 32 |
| 6. | TRIAL OBJECTIVES AND PURPOSE | 36 |
| 6.1. | Primary Objective | 36 |
| 6.2. | Secondary Objective | 36 |
| 6.3. | Exploratory Objectives | 36 |
| 6.4. | Safety Objective | 37 |
| 7. | INVESTIGATIONAL PLAN | 38 |
| 7.1. | Overall Trial Design | 38 |
| 7.2. | Number of Patients | 40 |
| 7.3. | Criteria for Trial Termination | 40 |
| 8. | SELECTION AND WITHDRAWAL OF PATIENTS | 41 |
| 8.1. | Patient Inclusion Criteria | 41 |
| 8.2. | Patient Exclusion Criteria | 41 |
| 8.3. | Patient Withdrawal Criteria | 43 |
| 9. | TREATMENT OF PATIENTS | 44 |
| 9.1. | Description of Trial Product | 44 |
| 9.2. | Prior and Concomitant Medications | 44 |

#### Protocol Version 7.0/Amendment 6/25 Jun 2020

| 9.2.1. | Prophylactic Administration of Prednisolone | 44 |
|---|---|---|
| 9.2.2. | Prohibited Medications | 45 |
| 9.2.3. | Vaccinations | 45 |
| 9.3. | Treatment Compliance | 46 |
| 9.4. | Randomization and Blinding | 46 |
| 10. | TRIAL PRODUCT MATERIALS AND MANAGEMENT | 47 |
| 10.1. | Trial Product | 47 |
| 10.2. | Trial Product Dose and Dose Justification | 47 |
| 10.3. | Trial Product Packaging and Labeling. | 47 |
| 10.4. | Trial Product Storage and Destruction. | 47 |
| 10.5. | Trial Product Preparation | 48 |
| 10.6. | Trial Product Administration | 48 |
| 10.7. | Dose Adjustment Criteria | 48 |
| 10.8. | Trial Product Accountability | 48 |
| 10.9. | Trial Product Handling and Disposal | 48 |
| 11. | ASSESSMENT OF EFFICACY | 50 |
| 11.1. | Developmental Milestones | 50 |
| 11.2. | Motor Function Tests | 51 |
| 11.2.1. | World Health Organization Multicentre Growth Reference Milestones | 51 |
| 11.2.2. | Bayley Scales for Infant and Toddler Development/Developmental Milestones | 51 |
| 11.2.3. | CHOP INTEND | 52 |
| 11.3. | Video Evidence | 52 |
| 12. | ASSESSMENT OF SAFETY | 54 |
| 12.1. | Safety Parameters | 54 |
| 12.1.1. | Demographic/Medical History | 54 |
| 12.1.2. | Physical Examinations | 54 |
| 12.1.3. | Vital Signs/Weight and Length | 55 |
| 12.1.4. | Electrocardiogram | 55 |
| 12.1.5. | Echocardiogram | 55 |
| 12.1.6. | Continuous ECG Recordings. | 56 |
| 12.1.7. | Pulmonary Examinations | 56 |

| Investigational Product: AVXS-101 | | ocol Version 7.0/Amendment 6/25 Jun 2020 |
|---|---|---|
| 12.1.8. | Swallowing Test | 56 |
| 12.1.9. | Photographs of Infusion Site | 56 |
| 12.1.10. | Laboratory Assessments | 57 |
| 13. | ADVERSE AND SERIOUS ADVERSE EVEN | ΓS62 |
| 13.1. | Definition of Adverse Events | 62 |
| 13.1.1. | Adverse Event | 62 |
| 13.1.2. | Serious Adverse Event | 62 |
| 13.1.3. | Adverse Events of Special Interest | 63 |
| 13.2. | Relationship to Trial Drug | 63 |
| 13.3. | Recording Adverse Events | 63 |
| 13.4. | Reporting Adverse Events | 64 |
| 13.5. | Expedited Safety Reporting to Regulatory Author | orities64 |
| 14. | STATISTICS | 65 |
| 14.1. | Data Analysis | 65 |
| 14.1.1. | Trial Endpoints and Populations | 65 |
| 14.2. | Sample Size Calculation | 68 |
| 14.3. | Efficacy Analysis | 70 |
| 14.3.1. | General Considerations | 70 |
| 14.3.2. | Primary and Secondary Efficacy Analysis | 70 |
| 14.4. | Safety Analysis | 71 |
| 14.4.1. | Hy's Law Criteria | 71 |
| 15. | DATA SAFETY MONITORING BOARD/DAT<br>COMMITTEE | |
| 16. | DIRECT ACCESS TO SOURCE DATA/DOCU | MENTS73 |
| 16.1. | Trial Monitoring | 73 |
| 16.2. | Audits and Inspections | 73 |
| 16.3. | Institutional Biosafety Committee | 74 |
| 16.4. | Institutional Review Board/Independent Ethics C | Committee74 |
| 17. | QUALITY CONTROL AND QUALITY ASSU | RANCE75 |
| 18. | ETHICS | 76 |
| 18.1. | Ethics Review | 76 |
| 18.2. | Ethical Conduct of the Trial | 76 |

| Investigation | nal Product: AVXS-101 Protocol Version 7.0/Amendment 6/25 J | un 2020 |
|---|---|---|
| 18.3. | Written Informed Consent | 76 |
| 19. | DATA HANDLING AND RECORDKEEPING | 78 |
| 19.1. | Electronic Case Report Forms | 78 |
| 19.2. | Inspection of Records | 78 |
| 19.3. | Retention of Records | 78 |
| 20. | PUBLICATION POLICY | 79 |
| 21. | LIST OF REFERENCES | 80 |
| 22. | APPENDICES | 84 |
| APPENDI | X 1. SCHEDULE OF ASSESSMENTS | 84 |
| APPENDI | X 2. POST-MORTEM TISSUE AND ORGAN COLLECTION PLAN | 88 |
| APPENDI | X 3. BAYLEY SCALES OF INFANT AND TODDLER DEVELOPMENT (VERSION 3) | 90 |
| APPENDI | X 4. PERFORMANCE CRITERIA FOR BAYLEY SCALES INFANT AND TODDLER DEVELOPMENT (VERSION 3) DEVELOPMENTAL MILESTONES | 115 |
| A DDENINI | X 5. PERFORMANCE CRITERIA FOR WORLD HEALTH | 113 |
| AITENDI | ORGANIZATION (WHO) DEVELOPMENTAL MILESTONES | 116 |
| APPENDI | X 6. CHOP INTEND | 117 |
| APPENDI | X 7. DECLARATION OF HELSINKI: ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS | 120 |
| APPENDI | X 8. SUMMARY OF CHANGES | 126 |
| | LIST OF TABLES | |
| Table 1: | Spinal Muscular Atrophy Classification | 25 |
| Table 2: | Investigational Product | 44 |
| Table 3: | Total Blood Volume | 57 |
| Table 4: | Common Terminology Criteria for Adverse Events | 62 |
| Table 5: | Tissue Sample for Analysis | 88 |
| | LIST OF FIGURES | |
| Figure 1: | Kaplan-Meier Survival Curves and Survival Probabilities for SMA Types 1, 2, and 3 | 26 |
| Figure 2: | Trial Results, Including Staining of Transduced Spinal Motor Neurons, SMN Expression Levels, Righting Ability, and Weight and Survival Curves | |
| Figure 3: | Body Mass of Treated and Control Mice Showed No Difference | |

| PRO-747 Vers | sion7.0 Generated 22 Sep 2020 08 | 3:42 PM CEST Effective Date: 03 Jul 2020 08:04 PM CEST |
|---|---|---|
| AveXis, Inc. | | AVXS-101-CL-302 |
| Investigatio | nal Product: AVXS-101 | Protocol Version 7.0/Amendment 6/25 Jun 2020 |
| Figure 4: | Trial Design | 39 |


# 4. LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

The following abbreviations and specialist terms are used in this trial protocol.

| Abbreviation or Specialist Term | Explanation |
|---|---|
| AAV | Adeno-associated virus |
| AAV9 | Adeno-associated virus serotype 9 |
| ADL | Activities of daily living |
| AE | Adverse event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| APTT | Activated partial thromboplastin time |
| ASO | Antisense oligonucleotide |
| AST | Aspartate aminotransferase |
| BSIDv03 | Bayley Scales of Infant and Toddler Development, version 3 |
| BUN | Blood urea nitrogen |
| СВ | Chicken-β-actin-hybrid |
| cGMP | Current Good Manufacturing Practice |
| CHOP INTEND | Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders |
| СК | Creatine kinase |
| СК-МВ | Creatinine kinase-muscle/brain |
| CMV | Cytomegalovirus |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ddPCR | Droplet digital polymerase chain reaction |
| DMC | Data Monitoring Committee |
| DRG | Dorsal root ganglia |
| Day 1 | First 24-hour interval after the start of gene replacement therapy infusion |
| Day -1 | 24-hour interval prior to the start of gene replacement therapy infusion |

Investigational Product: AVXS-101


| Abbreviation or Specialist Term | Explanation |
|---|---|
| DSMB | Data Safety Monitoring Board |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-linked immunosorbent assay |
| ELISpot | Enzyme-linked immunospot |
| FVB | Friend virus B-type |
| GCP | Good Clinical Practice |
| GFP | Green fluorescent protein |
| GGT | Gamma glutamyl transferase |
| GLP | Good Laboratory Practice |
| HEENT | Head, eyes, ears, nose, and throat |
| HIV | Human immunodeficiency virus |
| ICD-10 code | International Statistical Classification of Diseases and Related Health Problems |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IRB | Institutional Review Board |
| ITR | Inverted terminal repeat |
| ITT | Intent-to-treat |
| IV | Intravenous |
| LFE | Liver function enzymes |
| LFT | Liver function test |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MGRS | Multicenter Growth Reference Study |
| NHP | Non-human primates |

Investigational Product: AVXS-101


| Abbreviation or Specialist Term | Explanation |
|---|---|
| NOAEL | No observable adverse effect level |
| PBMC | Peripheral blood mononuclear cells |
| PICU | Pediatric intensive care unit |
| PNCR | Pediatric Neuromuscular Clinical Research Network |
| RSV | Respiratory syncytial virus |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| Sc | Self-complementary |
| scAAV | Self-complementary adeno-associated virus |
| scAAV9.CB.SMN | Self-complementary adeno-associated virus serotype 9 chicken-β-actin-hybrid survival motor neuron |
| SMA | Spinal muscular atrophy |
| SMN | Survival motor neuron |
| SMN1 | Survival motor neuron 1 gene |
| SMN2 | Survival motor neuron 2 gene |
| SoA | Schedule of Assessments |
| SUSAR | Suspected unexpected serious adverse reaction |
| TBL | Total bilirubin |
| ULN | Upper limits of normal |
| US | United States |
| vg/kg | Vector genome per kilogram |
| WBC | White blood cell |
| WHO | World Health Organization |
| WT | Wild type |


#### 5. INTRODUCTION

Trial AVXS-101-CL-302 is a pivotal Phase 3 clinical gene therapy trial investigating the efficacy and safety of a single intravenous (IV) infusion of AVXS-101 in 30 patients with Type 1 spinal muscular atrophy (SMA) with 1 or 2 copies of survival motor neuron 2 gene (SMN2). The survival motor neuron (SMN) gene will be transferred using self-complementary adenoassociated virus (scAAV) Type 9 under control of the chicken-β-actin hybrid promoter. Pre-clinical studies have demonstrated survival of the SMNΔ7 mouse model for SMA from a median of 15.5 days to over 1 year, following IV delivery to the peripheral vein. Additionally, preliminary results from a completed Phase 1 clinical trial (AVXS-101-CL-101) of AVXS-101 in SMA Type 1 patients demonstrates broad improvements in survival, motor function, pulmonary function, and nutritional function (Section 5.4).

# 5.1. Background

Spinal muscular atrophy is a neurogenetic disorder caused by a loss or mutation in the survival motor neuron 1 gene (SMNI) on chromosome 5q13, which leads to reduced SMN protein levels and a selective dysfunction of motor neurons. Spinal muscular atrophy is an autosomal recessive, early childhood disease with an incidence of approximately 1: 10,000 live births [1]. Spinal muscular atrophy is the leading cause of infant mortality due to genetic diseases. Disease severity and clinical prognosis depends on the number of copies of survival motor neuron 2 gene (SMN2). In its most common and severe form (Type 1), hypotonia and progressive weakness are recognized in the first few months of life, leading to diagnosis before 6 months of age and early death due to respiratory failure before 2 years of age. Motor neuron loss in SMA Type 1 is profound in the early post-natal period (or may even start in the prenatal period), whereas motor neurons in SMA Type 2 and Type 3 patients adapt and compensate during development and many will persist into adult life. The findings from various neurophysiological and animal studies have shown an early loss of motor neurons in the embryonic and early post-natal periods [2,3,4]. From a clinical perspective, these findings emphasize the importance of first targeting the SMA Type 1 group for gene transfer of SMN2 in hopes of rescuing neurons at this critical stage. The goal in continuing the development plan for AVXS-101 is to modify the SMA Type 1 phenotype, which will hopefully lead to a milder disease course and prolonged survival as seen in SMA Type 2 and Type 3 patients.

Therapeutic efforts in SMA have focused on the potential for small molecules to increase SMN protein levels. These include deacetylase inhibitors, such as, valproic acid, sodium butyrate, phenylbutyrate, and trichostatin A. These agents activate the *SMN2* promoter, resulting in increased full-length SMN protein in SMA animal models [5,6]; however, clinical studies employing several of these agents, most notably phenylbutyrate, valproic acid, and hydroxyurea, have not resulted in clinical benefit [7,8]. In the United States, the Food and Drug Administration (FDA) recently approved nusinersen, an antisense oligonucleotide (ASO) drug designed to increase the production of the SMN protein by modulating the splicing of the *SMN2* gene, thereby compensating for the underlying genetic defect. Clinical studies have shown some modest promise in improving motor function; however, the treatment must be administered indefinitely on a quarterly basis via intrathecal injection, requires a lengthy induction period prior to effectiveness, and has safety considerations that require clinical monitoring. A single-dose IV administration trial of AVXS-101 will provide information on the potential that

Investigational Product: AVXS-101


gene transfer has in treating SMA Type 1 patients and will hopefully show promise for success in modifying the disease prognosis.

This is a single-dose trial that will include up to 30 Type 1 patients with 1 or 2 copies of *SMN2*. The rationale for IV dosing is based upon the need for rapid, systemic impact given the severity of the disease in SMA Type 1 and its potential impact on systems outside of the central nervous system such as the peripheral and autonomic nervous systems, heart, pancreas and gastrointestinal tract.

## **5.2.** Rationale for Gene Transfer to SMA Type 1 Patients

Patients with SMA Type 1 have been chosen as the target population for this gene therapy trial based on studies of the natural history of this disease. The classification of SMA is shown below (Table 1) in which SMA Types 0 to 4 are described. Spinal muscular atrophy is conventionally classified into 4 phenotypes on the basis of age at onset and highest motor function achieved, with an additional phenotype (Type 0) to describe the severe forms of antenatal-onset SMA [9].

Table 1: Spinal Muscular Atrophy Classification

| Type | Age at S | ymptom Onset | Maximum Motor<br>Function | Life Expectancy | SMN2 Copy No. |
|---|---|---|---|---|---|
| 0 | Fetal | | Nil | Days – Weeks | 1 |
| 1 | < 6 Months | 1A: B-2 Weeks<br>1B: < 3 months<br>1C: > 3 months | Never sits | < 2 years | 1, 2, 3 |
| 2 | 6 – 18 Months | | Never walks | 20 – 40 years | 2, <b>3</b> , 4 |
| 3 | 1.5 – 10 Years | 3A: < 3 Years<br>3B: > 3 Years | Walks, regression | Normal | 3, 4, 5 |
| 4 | > 35 Years | | Slow decline | Normal | 4, 5 |

Source: Adapted from Kolb 2011[10] SMN2 = survival motor neuron 2 gene

**bold** = predominant *SMN2* copy number that defines the SMA Type, the other copy numbers represent a small percentage of the designated SMA Type.

Spinal muscular atrophy Type 1 patients, by definition, never attain independent sitting and have hypotonia within the first 6 months of life. Spinal muscular atrophy Type 1 is the leading genetic cause of infant death with an onset at  $\leq 6$  months of age (Table 1). In contrast, SMA Type 2 manifests within the first 18 months, and children afflicted with this condition are able to maintain sitting unassisted but never walk independently. Spinal muscular atrophy Type 3 patients attain the ability to walk unaided (Type 3a have onset 18 months to 3 years of age; Type 3b have onset  $\geq$  3 years of age). Spinal muscular atrophy Type 4 is an adult onset disease. The genetic cause for SMA is well established and is intimately involved with one's prognosis. All forms of SMA are autosomal recessive in inheritance and are caused by deletions or mutations of the *SMN1* gene.

Humans also carry a second nearly identical copy of the *SMN1* gene called *SMN2* [11]. Both the *SMN1* and *SMN2* genes express SMN protein; however, the amount of functional full-length protein produced by *SMN2* is only 10 to 15% of that produced by *SMN1* [11,12,13]. Although

Investigational Product: AVXS-101


SMN2 cannot completely compensate for the loss of the SMN1 gene, patients with milder forms of SMA generally have higher SMN2 copy numbers [14,15]. Quantitative analysis of SMN2 copies in 375 patients with Type 1, 2, or 3 SMA showed a significant correlation between SMN2 copy number and SMA Type, as well as, duration of survival. In a large early trial by Feldkotter et al 2002 [16], 2 copies of SMN2 was 97% predictive for developing SMA Type 1, 3 copies of SMN2 was 83% predictive for developing SMA Type 2, and 4 copies of SMN2 was 84% predictive of SMA Type 3. As these percentages do not reflect the possible impact of modifier mutations such as that described by Prior et al 2009 [17], they may understate the relationship between copy number (in the absence of a genetic modifier) and clinical phenotype. Among 113 patients with Type 1 SMA, 9 with 1 SMN2 copy lived < 11 months, 88/94 with 2 SMN2 copies lived < 21 months, and 8/10 with 3 SMN2 copies lived 33 to 66 months. Even more refined data describing this relationship has been generated and has also influenced our choice of the trial target group.

The severity of SMA Type 1 is demonstrated by prognosis as illustrated in Kaplan-Meier survival curves shown in Figure 1.

Figure 1: Kaplan-Meier Survival Curves and Survival Probabilities for SMA
Types 1, 2, and 3



n = number of patients Source: Farrar 2013 [18]

In Figure 1, the relative stability of the clinical course of SMA Type 2 and Type 3 is dramatically illustrated. Perhaps most importantly, these findings show that outcome differences are related to the number of *SMN2* copies that enable motor neurons to adapt and compensate during the growth of the child and persist into adult life. This contrasts with SMA Type 1 where motor neuron loss is profound in the early post-natal period (or may even start in the prenatal period, especially for SMA Type 1 patients presenting in first 3 months of life). The findings in Figure 1 confirm other pieces of evidence from neurophysiological studies and animal studies that also show early loss of motor neurons in the embryonic and early post-natal periods [2,3,4].

Investigational Product: AVXS-101


There is reason to believe that there are few safety issues to be concerned about when targeting the SMA Type 1 group in this gene therapy clinical trial. Overexpression of SMN protein has been shown to be well tolerated in both mice and non-human primates, and in humans, a high copy number of *SMN2* poses no risk (as seen in Type 2, 3, and 4 patients who have high *SMN2* copy number), allowing for use of robust, ubiquitous expression systems (like the chicken β-actin-hybrid (CB)-promoter) to ensure sustained, high-level SMN gene expression. Additionally, it is important to point out that recombinant scAAV can be employed for this trial because of the small size of the SMN gene. This enables efficient packaging and allows for efficient gene transfer with lower viral titers (a safety consideration), compared with prototypical single-stranded AAV vectors.

Recent studies using self-complementary adeno-associated virus serotype 9 chicken-β-actin-hybrid survival motor neuron (scAAV9.CB.SMN) show a robust post-natal rescue of SMNΔ7 mice with correction of motor function, neuromuscular electrophysiology and survival after a 1-time delivery of vector [19]. Intravenous scAAV9 is able to transduce neurons, muscle and vascular endothelium, all of which have been proposed as target cells for SMA treatment.

#### **5.3.** Nonclinical Studies

A mouse model was developed by the after a generation of evaluating various transgenic permutations. It was found that the double transgenic, referred to as the SMN $\Delta$ 7 mouse, provided the most suitable model to trial gene transfer [20]. Studies have shown that injecting  $5 \times 10^{11}$  viral genomes of performed in the scAAV9.CB.SMN into the facial vein on post-natal Day 1 rescues mice in the SMNΔ7 mouse model [19]. Figure 2 shows the results of these studies, including staining of transduced spinal motor neurons, SMN protein expression levels, righting ability, and weight and survival curves. Approximately  $42 \pm 2\%$  of lumbar spinal motor neurons were transduced in scAAV9.CB.GFP treated mice. SMN transduction was shown by real time polymerase chain reaction (RT-PCR) in the mice. Green fluorescent protein (GFP) transduction was observed by microscopy. Both constructs were in adeno-associated virus serotype 9 (AAV9) and had transduction of motor neurons. SMN protein levels were increased as well, in brain, spinal cord, and muscle of scAAV9.CB.SMN-treated animals, compared to untreated SMNΔ7 mice (although lower than wild type [WT] controls). SMNΔ7 animals treated with either scAAV9.CB.SMN or scAAV9.CB.GFP on post-natal Day 1 (P1) were assessed for their righting ability and were compared to WT control mice and untreated mice. Wild type controls could right themselves quickly, whereas the SMN- and GFP-treated SMA animals showed difficulty at P5; however, by P13, 90% of SMN-treated animals could right themselves compared with 20% of GFP-treated controls and 0% of untreated SMA animals. At P18, SMN-treated animals were larger than GFP-treated animals, but smaller than WT controls. Locomotive ability of the SMN-treated mice was nearly identical to WT controls, as assayed by open field testing and wheel running.

Survival of SMN-treated SMNΔ7 animals compared with GFP-treated SMNΔ7 animals was significantly improved. No GFP-treated control animals survived past P22 and had a median life span of 15.5 days. The weights of GFP mice peaked at P10 and then precipitously declined until death, while SMN mice showed a steady weight gain until around P40 with it stabilizing at 17 g (about half the weight of WT controls). The smaller size of corrected animals is likely related to the tropism and incomplete transduction of scAAV9, resulting in a 'chimeric' animal in which

Investigational Product: AVXS-101


some cells were not transduced. Additionally, the smaller size suggests an embryonic role for SMN protein. Most remarkably, SMN-treated mice survived well past 250 days of age.

Figure 2: Trial Results, Including Staining of Transduced Spinal Motor Neurons, SMN Expression Levels, Righting Ability, and Weight and Survival Curves



Source: Foust 2010 [19]

CNS = central nervous system; GFP = green fluorescent protein; SMN = survival motor neuron; WT = wild type

- a. Shows transduced motor neurons in lumbar spinal cord
- **b.** Western Blots of SMN expression in CNS and muscle
- c. Improved righting ability of SMN-treated-similar to WT controls by post-natal Day 13 (P13)
- **d.** SMN-treated are larger than GFP-treated at P18
- e. Survival of SMN-treated markedly improved compared to GFP-treated
- f. Body weight increased in SMN-treated vs GFP

Toxicology biodistribution studies were generated by the **Section 1** [data on file]. In these non-Good Laboratory Practice (non-GLP) studies, 24 mice and 4 non-human primates

Investigational Product: AVXS-101


(NHPs) were injected, by way of vascular delivery, with AVXS-101. To assess toxicity and safety, AVXS-101 was injected into post-natal Day 1 (P1) wild type Friend Virus B-Type (FVB) mice with either vehicle (3 males/6 females) or 3.3 × 10<sup>14</sup> vector genome per kilogram (vg/kg) of AVXS-101 (previously known as scAAV9.CB.SMN (6 males/9 females) via the facial temporal vein. This dose was previously shown to be most efficacious in the SMNΔ7 mouse model [19]. P1 mice were used in anticipation of simulating potential clinical studies in infants. All mice survived the injection procedure and the initial 24-hour observation period without any signs of distress or weight loss. Body mass was measured and hands-on observations were performed weekly for the remainder of the trial; neither revealed any difference between control and treated cohorts (Figure 3).



Figure 3: Body Mass of Treated and Control Mice Showed No Difference

At 60, 90, and 180 days post-injection, blood from the mice was collected for hematology studies including complete blood counts with differentials. At 90, 120, and 180 days post-injection, blood was collected for clinical chemistries assessment (alanine amino transferase [ALT], aspartate amino transferase [AST], alkaline phosphatase, creatinine, blood urea nitrogen [BUN], electrolytes, and creatine kinase [CK]). For histopathology, 13 mice were necropsied at 120 days post-injection and 8 mice at 180 days. There were no clinically significant results observed during from the hematology, clinical chemistry, and histopathology portions of the trial and trends of both groups were comparable. Of note, no significant lesions were present in any brain or spinal cord sections, although, the sections were frozen and thicker than 5 microns which may obscure subtle changes in cellular morphology.

In the safety trial for the 4 male cynomolgus macaques, animals were injected at 90 days of age to closely mimic the likely age of administration of treatment in SMA Type 1 infants. The AVXS-101 vector was administered 1 time by catheterization of the saphenous vein with a dose of  $6.7 \times 10^{13}$  vg/kg, which corresponds to the lowest dose tested for which SMN $\Delta$ 7 mice showed a significant increase of survival. Animals were followed for 6 months until they were sacrificed at approximately 9 months of age. No adverse effects were seen, and all clinical chemistries were normal. T-cell immune response was tested using enzyme-linked immunospot (ELISpot)

Investigational Product: AVXS-101


in peripheral blood mononuclear cells (PBMCs), and all were negative at 6 months post-injection.

In these non-GLP studies, the serum chemistry and hematology data were unremarkable as was the histopathology assessment. The NHPs mounted appropriate immune responses to capsid (but not to transgene), with very high transgene expression persisting at 6 months post-injection. In conclusion, these studies provide strong evidence that systemically-delivered scAAV9.CB.SMN is safe and well tolerated, even at the high doses required for penetration of the blood-brain barrier [19].

When newborn FVB mice were given a single IV injection of AVXS-101 at levels up to  $3.3 \times 10^{14} \, \text{vg/kg}$  on Day 1, there was neither test article-related mortality nor evidence of toxicity seen at timepoints up to 24 weeks after administration. Treatment-related decreases in mean body weight and mean body weight gain, as well as lower activated partial thromboplastin time (APTT) values, were mild effects of treatment, but did not result in toxicity. Activity of AVXS-101 was demonstrated by the biodistribution and the presence of a specific transgene ribonucleic acid expression in brain and spinal cord, the main targeted therapeutic tissues. Low levels of antibodies to the AAV9 capsid were found after 12 and 24 weeks in males and females given  $3.3 \times 10^{14} \, \text{vg/kg}$  (Group 3). No alteration was observed in clinical pathology and histopathology analyses.

As part of the preclinical development of AVXS-101 for intrathecal delivery, an exploratory non-GLP biodistribution and safety study was performed in cynomolgus monkeys (Macaca fascicularis) to evaluate the transduction efficiency and safety of intrathecally administered AVXS-101 at a dose of 3 x 10<sup>13</sup> vg/animal alone and in combination with 2 iohexol-based contrast agents. All 12 animals on study survived and were euthanized 2 weeks post-injection with no clinical evidence of toxicity. However, inflammation of the dorsal root ganglia (DRG) was noted during histopathology evaluation of select tissues. The inflammation was characterized by minimal to marked infiltration of mononuclear inflammatory cells, primarily lymphocytes, into the cervical, thoracic, lumbar, and sacral DRGs and associated nerves. Minimal inflammation was associated with scattered infiltrates or small aggregates of mononuclear cells in the DRG, without evidence of neuronal necrosis. With mild to marked inflammation, aggregates to sheets of mononuclear cells were present, along with neuronal satellitosis, neuronal necrosis, or neuronal loss with rare mineralization. Inflammation was observed in ganglia from all examined levels, but incidence and severity were generally greater in the sacral DRG. Moderate to marked inflammation was only observed in the sacral DRG of 2 of the 12 animals on study. The animals were not administered corticosteroids.

The DRG was not identified as a target organ of toxicity in previous AVXS-101 studies conducted in mice (ICV route of administration) or cynomolgus monkeys (IV or IT routes of administration). However, similar findings have been reported after administration of an AAV9 vectors in monkeys and minipigs (20, 21).

In pivotal GLP-compliant 3-month mouse toxicology studies, the main target organs of toxicity were the heart and liver. Following IV infusion in the mouse, vector and transgene were widely distributed with the highest expression generally observed in heart and liver, and substantial expression in the brain and spinal cord. AVXS-101-related findings in the ventricles of the heart were comprised of dose-related inflammation, edema and fibrosis, and in the atrium,

Investigational Product: AVXS-101


inflammation and thrombosis. Liver findings were comprised on hepatocellular hypertrophy, Kupffer cell activation, and scattered hepatocellular necrosis. A no observable adverse effect level (NOAEL) was not identified for AVXS-101-related heart and liver findings in the mouse, and the maximum tolerated dose was defined as  $1.5 \times 10^{14}$  vg/kg, providing a safety margin of approximately 1.4-fold relative to the recommended therapeutic dose of  $1.1 \times 10^{14}$  vg/kg. The translatability of the observed findings in mice to primates is not known at this time.

#### **5.4.** Clinical Studies

First-in-human trial AVXS-101-CL-101 is a completed 2-year trial which evaluated the efficacy and safety of AVXS-101 in 15 SMA Type 1 patients with 2 copies of SMN2. All patients have received a single IV dose of AVXS-101 in 2 cohorts: Cohort 1 (n = 3) received  $6.7 \times 10^{13} \text{ vg/kg}$  and Cohort 2 (n = 12) received  $2.0 \times 10^{14} \text{ vg/kg}$  (proposed therapeutic dose). After the End of Trial visit, patients were invited to participate in a long term follow up study conducted under a separate protocol.

- Based on data obtained in Study AVXS 101-CL-101, the following conclusions can be made regarding the efficacy of AVXS 101:
- AVXS 101 administration had a positive effect on survival. Twenty-four months after
  dosing, all 15 patients were alive and free of permanent ventilation 24 months after
  dosing and all Cohort 2 patients had survived free of permanent ventilation, a statistically
  significant difference compared with the natural history rate of 8% reported by Finkel et
  al 2014 [23].
- Based on independent video reviews, developmental milestones were achieved and maintained over time.
  - o In Cohort 2, 11 patients (91.7%) could hold their head erect without support for ≥ 3 seconds and sit with support, 9 patients (75.0%) were able to sit without support for ≥ 30 seconds, and 2 patients each (16.7% each) were able to stand with assistance, stand alone, walk with assistance, and walk alone
- The improvements in Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) scores from baseline in both cohorts were sustained over time.
- Nearly all Cohort 2 patients (11/12, 91.7%) achieved a score ≥ 50 on the CHOP INTEND, approximating the range of scores for Type 2 SMA children reported in the Pediatric Neuromuscular Clinical Research Network (PNCR) study [23].
- Other clinically meaningful milestones were maintained 24 months after AVXS-101 infusion:
  - Of the 7 patients in Cohort 2 who did not require non-oral nutrition prior to AVXS-101 dosing, 5 (71.4%) maintained the ability to thrive
  - Eleven Cohort 2 patients (91.7%) were still able to swallow effectively enough to feed orally
  - O Seven of 15 patients (46.7%) remained independent of ventilatory support


#### **5.5.** Risks

A full understanding of all the risks associated with AVXS-101 is not known at this time. Potential risks of AVXS-101 are discussed below and further details are provided in the Investigator's Brochure [25].

Patients could experience an allergic response to AVXS-101. Patients could also develop an immune response to the AAV9 viral vector, which could prevent future use of gene transfers using this vector.

Some mice affected with a form of SMA Type 1 that were treated with the study vector developed localized vascular necrosis around the ear called necrotic pinna. This is believed to be unrelated to the vector, and likely related to an underlying defect that has been observed to occur in several SMA mouse models [26]. The relevance to humans with SMA is unknown.

Respiratory tract infections in neonates are very common in the general pediatric population [27]. In one study, an estimated 338 million new episodes of respiratory syncytial virus (RSV) - associated acute lower respiratory infections occurred worldwide in children younger than 5 years, with at least 34 million episodes necessitating hospital admission [28]. RSV is the primary cause of hospitalization for respiratory tract infection in young children [29]. It would not be unexpected that infants enrolled in the AVXS-101 gene replacement therapy trials might have similar incidences of respiratory infections due to these pathogens.

Patients must be clinically stable before AVXS-101 dosing. Clinical signs or symptoms of infection should not be evident at the time of AVXS-101 administration. Vaccinations, including palivizumab prophylaxis that can prevent RSV infections [30], are also recommended [31] and should be up to date. Added caution is advised regarding the timing of AVXS-101 administration in the presence of prodrome or resolving viral illness. In the event of a severe viral respiratory infection, the Investigator should be aware of the possibility of adrenal insufficiency in the presence of systemic immune response which may require longer glucocorticosteroid support at increasing doses to effectively manage the patient and prevent serious complications.

Some mice affected with SMA Type 1 that were treated with AVXS-101 experienced liver findings comprised of hepatocellular hypertrophy, Kupffer cell activation, and scattered hepatocellular necrosis.

Adverse events (AEs) of increased transaminases (ALT increased, AST increased, and transaminase increased) were reported as related to AVXS-101 in clinical studies. The underlying cause of the transaminase elevations is not known; though, may be related to an immune response to AAV9, as indicated by the response to prednisolone. Though these AEs can be serious, in most cases they were clinically asymptomatic, did not meet criteria for Hy's law (Section 14.4.1), did not exhibit clinically relevant increases in bilirubin, and generally resolved with prednisolone treatment. A case of acute liver failure (suspected unexpected serious adverse reaction [SUSAR]) was reported in the US Managed Access Program with AVXS-101. A 6-month-old male concurrently receiving nusinersen with elevations of AST and ALT of > 3 x the upper limit of normal (ULN) before treatment with AVXS-101 developed acute liver failure approximately 51 days post AVXS-101 dosing. The patient recovered with additional steroid therapy.

Investigational Product: AVXS-101


Nonclinical cardiovascular toxicity findings that could potentially be relevant to the clinical use of AVXS-101 have been reported in 2 mouse toxicology studies of AVXS-101. Similar findings were reported in both studies. Findings in the ventricles of the heart were comprised of inflammation, edema and fibrosis. Primary findings in the atrium of the heart were thrombosis and inflammation. The underlying mechanism of these findings and the translatability of the observed findings in mice to primates are not known at this time.

The available clinical cardiovascular safety data have not provided evidence for a cardiovascular safety problem in humans. As of the last update to the IB, there have been no cardiovascular AEs that have been judged to be related to AVXS-101 in the clinical studies. There have been no persistent clinically significant electrocardiogram (ECG) changes. In Study AVXS-101-CL-303, a Phase 3 open-label single-dose study in patients with one or two copies of SMN2, elevated CK-MB was reported for one patient, but this TEAE was determined by the Investigator to be unrelated to AVXS-101 administration. There have been no AEs reported for troponin-I. In Study AVXS-101-CL-101, there were minor transient increases in troponin-I at the proposed therapeutic dose in Cohort 2 with no associated clinical sequelae. None of the elevations in cardiac troponin-I observed during the study were considered clinically significant by the investigator. Small mean troponin elevations were minimally apparent during the first two months post-dose. Other troponin elevations appeared to be sporadic. By the end of the study all values had either returned to within the normal range or no longer met the pre-defined criterion for potential clinical significance. The autopsy report from Study AVXS-101-CL-303 patient, whose death was unrelated to AVXS-101, indicates that the heart was macroscopically and microscopically normal, with sections of the heart having no pathologic diagnosis. While the clinical significance of the transiently elevated troponin-I levels is unknown, it is recommended that troponin-I be monitored for the first 3 months following dosing.

A transient decrease in platelet counts has been observed in Studies AVXS-101-CL-101, AVXS-101-CL-303, and AVXS-101-CL-102 typically at Day 7. The majority of values remained above the lower limit of normal. Decreases were clinically asymptomatic and transient.

Preclinical data indicate that in most cases, DNA delivered by recombinant AAV vectors predominantly persists as extrachromosomal elements (episomes) rather than integrating into host cell genomes [32]. Although AVXS-101 is also not anticipated to integrate into the host cell genome as described above, the long-term consequences of administering AAV viral vectors to humans are not yet fully understood. This is in contrast to wild-type AAV, also non-pathogenic, which has the ability to stably integrate into the host cell genome at a specific site (designated AAVS1) in the human chromosome 19 [33, 34]. Since the AVXS-101 product uses AAV9 with all of the wild-type DNA removed from the capsids, except for the Inverted Terminal Repeats, the potential risk of incorporation of AVXS-101 into the patient chromosomal DNA is thought to be significantly reduced.

There are conflicting reports that integration of the wild-type AAV2 genome is associated with induction of hepatocellular carcinoma in a small subset of patients; however, there are several studies with evidence to contradict these claims including: a) AAV2 has infected approximately 90% of the human population, b) AAV2 has been shown to possess anticancer activity, c) epidemiological evidence suggests that AAV2 infection plays a protective role against cervical carcinoma, and d) AAV serotypes including recombinant AAV2 and AAV9 have been or are

Investigational Product: AVXS-101


currently used in 162 clinical trials to date in which no cancer of any type has been observed or reported. For a review of the topic, see Srivastava and Carter, 2017 [35]. Further support for the extremely low potential incorporation into host chromosomal DNA comes from pre-clinical studies, which to date have not shown the development of cancer in treated animals including mice and non-human primates exposed to AVXS-101.

It is possible the AAV9 vector containing the SMN gene could interact with other viruses with which the patients come in contact, such as rhinoviruses, adenovirus, or herpes. If this happens, the AAV9 vector could form a virus that causes infection if the patient and cells for rescue, replication, and packaging are also exposed to wild-type AAV2. The rescue, replication, and packaging would stop; however, as the helper viruses, such as rhinoviruses, adenovirus, or herpes were cleared by the patient's immune system. This unlikely scenario has been studied. In cell culture, the rAAV genome can be rescued and replicated by superinfection with wtAAV and a helper virus; however, in vivo rescue experiments have failed to show rescue and replication [36], except in 1 case in which very large doses of wtAAV and adenovirus were administered in a particular setting [37]. Therefore, AAV9 interaction with other viruses to cause infection appears to be a minimal risk for AVXS-101.

Studies have shown that some vector can be excreted from the body for up to a few weeks after injection/infusion; this is called "viral shedding". Vector shedding can be found in the blood, urine, saliva, and stool for up to a few weeks following injection. The risks associated with the shed vector are not known at this time; however, because the vector is non-pathogenic and cannot replicate, it is believed that shed vector is unlikely to result in clinically significant adverse effects. Regardless, instructions should be provided to patient families and caregivers regarding use of protective gloves if/when coming into direct contact with patient bodily fluids and/or waste, as well as good hand-hygiene for a minimum of 4 weeks after the injection. Additionally, patients are prohibited from donating blood for 2 years following the vector injection.

Viral shedding is dependent on a variety of factors including the route of administration of the product, the tropism of the virus or bacteria, and the natural route of transmission and shedding of the parent virus or bacterium from which the product is derived. AveXis collected saliva, urine, and stool samples at weekly timepoints through Day 30 and then monthly timepoints through Month 18 after gene transfer during the AVXS-101-CL-101 clinical study from 5 patients for viral shedding analysis. This analysis detects the number of genome copies by ddPCR in the applicable shed samples.

AVXS-101 is detectable in the shed samples from Day 1 post injection. Clearance of AVXS-101 is primarily via the feces and the majority of the dose is cleared within 30 days of dose administration. While initially concentrated in stool, the amount of vector shed declines logarithmically. In stool, levels 10% to 30% of the initial concentration in the body were detectable at Day 1 post infusion. At Day 14 post-infusion one patient showed a peak concentration in stool of 280% of initial concentration in body. In contrast, 3 patients for whom data were available showed a concentration of <1% of initial concentration in body at Day 14 post infusion. These concentrations declined approximately 4 logs over 30 days post dose, and all patients had levels of AVXS-101 in stool below the ddPCR limit of quantitation by 60 days post dose. Concentrations of vector shed in saliva and urine are quite low and are below the
Investigational Product: AVXS-101


ddPCR limits of quantitation in the matrices within days post-dose. AVXS-101 concentrations representing 0.1% to 0.01% of the initial dose (concentration) into the patient are found in urine and saliva at Day 1 post infusion, after which concentrations fell below the limit of quantitation of the assay [data on file]. Shed AAV vectors have been previously shown not to be infectious in urine and saliva excreta [36]. Together, these data demonstrate rapid decline of shed vector quantities well below initial concentrations in patients treated with AVXS-101.

In an exploratory non-GLP study, inflammation of the DRG (characterized by infiltration of mononuclear inflammatory cells, along with neuronal satellitosis and neuronal necrosis or loss) was observed 14 days after cynomolgus monkeys were administered AVXS-101 intrathecally. Although the inflammation was observed in ganglia from all examined levels (cervical, thoracic, lumbar, and sacral), the incidence and severity were generally greater in the sacral DRG. Neuronal toxicity is therefore a potential risk following IT administration of AVXS-101. No steroids were administered in the animal study (Section 5.3).

A thorough review of the safety data from patients treated with AVXS-101 based on a data cutoff of 31 December 2019 did not identify any adverse events related to sensory changes. Nevertheless, study participants will be closely monitored for any clinical manifestations of a potential DRG involvement.

Finally, there are potential risks associated with intravenous dosing. There may be a pain at the site of the infusion as well as bruising surrounding the infusion site. Infections are also possible at the site of the infusion.

These results also strongly support further clinical investigation of the efficacy and safety of AVXS-101 in patients with presymptomatic SMA. Because SMA is a progressive neurodegenerative disease which involves the irreversible neurodegeneration and death of motor neurons beginning before the onset of clinical symptoms, administration of gene replacement therapy as early as possible is believed to be of substantial importance for preventing motor neuron loss, maximizing the opportunity for patients to experience meaningful benefits from this treatment. This hypothesis is supported by data from the AVXS-101-CL-101 clinical study, which has included observations of substantial benefits in survival, motor function, and developmental milestone achievements relative to natural history, which were particularly striking for several patients treated at younger ages. Based on the current available data, safety events that appear to be associated with AVXS-101 consist of transient liver enzyme elevations which have resolved following treatment with prednisolone. Considering this favorable developing safety profile together with the potential for highly meaningful clinical benefits of early treatment, the risk-benefit relationship strongly supports further clinical investigation of AVXS-101 in infants with presymptomatic SMA.

Taken together, results from the clinical and nonclinical studies support further clinical investigation of the efficacy and safety of AVXS-101 in patients with SMA.


#### 6. TRIAL OBJECTIVES AND PURPOSE

# 6.1. Primary Objective

The primary objective is to:

• Determine efficacy by demonstrating achievement of developmental milestone of sitting without support for at least 10 seconds up to 18 months of age as assessed by World Health Organization (WHO) Motor Developmental Milestones (Appendix 5) [38].

# 6.2. Secondary Objective

The secondary objective is to:

• Determine efficacy based on survival at 14 months of age. Survival is defined by the avoidance of combined endpoint of either (a) death or (b) permanent ventilation which is defined by tracheostomy or by the requirement of ≥ 16 hours of respiratory assistance per day (via non-invasive ventilatory support) for ≥ 14 consecutive days in the absence of an acute reversible illness, excluding perioperative ventilation. Permanent ventilation, so defined, is considered a surrogate for death.

# 6.3. Exploratory Objectives

For the following exploratory efficacy endpoints, a Responder will be defined as a patient who demonstrates achievement of the endpoint at any post-procedure visit up to and including the 18-month trial visit:

- Determine efficacy by demonstrating achievement of developmental milestone of ability to hold head erect without support as defined by BSIDv03 Gross Motor Subtest Item #4 (Appendix 3 and Appendix 4) [39]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to roll over as defined by BSIDv03 Gross Motor Subtest Item #20 (Appendix 3 and Appendix 4) [39]
- Determine the efficacy by demonstrating achievement of developmental milestone of functional independent sitting for at least 30 seconds as defined by BSIDv03 item #26, (Appendix 3 and Appendix 4) [39]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand with assistance for at least 2 seconds as defined by BSIDv03 Gross Motor Subtest Item #33 (Appendix 3 and Appendix 4) [39]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to crawl forwards on hands and knees for a distance of at least 5 feet as defined by BSIDv03 Gross Motor Subtest Item #34 (Appendix 3 and Appendix 4) [39]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to pull to standing as defined by BSIDv03 Gross Motor Subtest Item #35 (Appendix 3 and Appendix 4) [39]

Investigational Product: AVXS-101


- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk with assistance as defined by BSIDv03 Gross Motor Subtest Item #37 (Appendix 3 and Appendix 4)[39]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand alone for at least 3 seconds as defined by BSIDv03 Gross Motor Subtest Item #40 (Appendix 3 and Appendix 4)[39]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk at least 3 steps without support as defined by BSIDv03 Gross Motor Subtest Item #42 (Appendix 3 and Appendix 4)[39]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to crawl as defined by WHO Motor Developmental Milestones (Appendix 5) [38]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand with assistance as defined by WHO Motor Developmental Milestones (Appendix 5) [38]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to stand alone as defined by WHO Motor Developmental Milestones (Appendix 5) [38]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk with assistance as defined by WHO Motor Developmental Milestones (Appendix 5) [38]
- Determine efficacy by demonstrating achievement of developmental milestone of ability to walk alone as defined by WHO Motor Developmental Milestones (Appendix 5) [38]
- Determine efficacy by demonstrating improvement of motor function as determined by improvement in the fine and gross motor domain components of the BSIDv03 (Appendix 3) [39]
- Determine efficacy by demonstrating improvement of gross motor function as determined by improvement in CHOP INTEND score (Appendix 6)
- Determine the effect of AVXS-101 on the ability to remain independent of ventilator support, defined as requiring no daily ventilator support/usage at 18 months of age.
- Determine effect on the ability to thrive defined as achieving all of the following:
  - Does not receive nutrition through mechanical support (i.e., feeding tube)
  - Ability to tolerate thin liquids as demonstrated through a formal swallowing test
  - Maintains weight (> third percentile for age and gender)

# **6.4.** Safety Objective

The safety objective is to:

• Evaluate the safety of AVXS-101 in patients with SMA Type 1


# 7. INVESTIGATIONAL PLAN

# 7.1. Overall Trial Design

This is a Phase 3, open-label, single-arm, single-dose trial of AVXS-101 (gene replacement therapy) in patients with SMA Type 1 with 1 or 2 copies of SMN2. Thirty patients < 6 months (< 180 days) of age <u>at the time</u> of gene replacement therapy (Day 1) are planned to be enrolled. Babies who are in screening and meet eligibility criteria for the study when the enrollment target is met may be enrolled upon approval of the sponsor.

The trial includes 3 trial periods: screening, gene replacement therapy, and follow-up (Figure 4). During the screening period (Days –30 to –2), patients whose parent(s)/legal guardian(s) provide informed consent will undergo screening procedures to determine eligibility for trial enrollment. Patients who meet the entry criteria will enter the in-patient gene replacement therapy period (Day –1 to Day 3). On Day –1, patients will be admitted to the hospital for pre-treatment baseline procedures. On Day 1, patients will receive a 1-time intravenous (IV) infusion of the equivalent of AVXS-101 Cohort 2 dose received in the AVXS-101-CL-101 trial over approximately 60 minutes, dependent upon required total volume, and will undergo in-patient safety monitoring over the next 48 hours. Patients may be discharged 48 hours after gene replacement therapy, based on Investigator judgment. During the outpatient follow-up period (Days 4 to End of Trial at 18 months of age), patients will return at regularly scheduled intervals for efficacy and safety assessments until the patient reaches 18 months of age. Any missed visit should be rescheduled as soon as possible, but within the visit windows shown in the Schedule of Assessments (SoA).

After dosing, follow-up visits will be conducted according to the SoA (Appendix 1). All post-treatment visits will be relative to the date on which gene replacement therapy is administered until the patient is 14 months of age, after which all visits will be relative to the patient's date of birth. For the 14 and 18 months of age visits, the patient will return within 0 to 14 days **after** the date on which the patient reaches 14 and 18 months of age, respectively. The 18 months of age visit will also serve as the End of Trial visit. After the End of Trial visit, patients will be invited to participate in a long term follow up study conducted under a separate protocol. Patients who discontinue prematurely will also be invited to participate in the long-term follow-up study.

In the event of unforeseen catastrophe or other, serious situation (such as the COVID-19 pandemic) that occurs during the study, which limits or prevents on-site study visits, alternative methods of conducting study assessments may be implemented. Phone calls, virtual contacts (e.g. teleconsult) or visits by site staff/home nursing service to the participant's home depending on local regulations and capabilities, can replace on-site study visits, for the duration of the pandemic until it is safe for the participant to visit the site again. The process for obtaining remote informed consent must be followed in order to conduct these alternative study visits (Section 18.3).

Throughout the study, the scheduling of study visits should adhere to the overall study schedule and visit windows defined in the protocol. For each study visit, all study procedures and assessments should be performed or completed in accordance with the schedule of events. Local institutions or other alternatives may be utilized.

Investigational Product: AVXS-101


Importantly, in instances in which the final scheduled study visit is not possible to be conducted at the study site or the scheduling of the final scheduled study visit is at risk of delay due to travel restrictions or other circumstances, the final scheduled study visit should be performed all or in part remotely within the protocol-defined visit window. Critical data that pertain to the co-primary and co-secondary endpoints and other information such as adverse events, concomitant medications, use of feeding or ventilatory support, or other safety data that may be obtained remotely should be collected as part of the final study visit and within the protocol-defined visit window.

Procedures such as laboratory and other safety assessments that cannot be performed or obtained as part of a remote visit may be performed separately and preferably within the protocol-defined visit window.

Figure 4: Trial Design



Note: After the End of Trial visit at 18 months of age or at the time of early discontinuation patients will be invited to participate in a long term follow up study conducted under a separate protocol.

In an attempt to dampen the host immune response to the AAV derived therapy, all patients will receive prophylactic prednisolone at approximately 2 mg/kg/day (or an equivalent dose of another glucocorticoid if prednisolone is unavailable or if, in the opinion of the investigator, prednisolone is not tolerated [41]) on Day -1, Day 1, and Day 2, and then 1 mg/kg/day starting on Day 3 and until at least 30 days post-AVXS-101 infusion. After 30 days post-AVXS-101 infusion, the dose of prednisolone can be tapered for patients whose gamma glutamyl transferase (GGT), ALT values, and AST values are below the threshold of 2 × ULN in accordance with the

All post-treatment visits will be relative to the date on which gene replacement therapy ("dose") is administered until the patient is 14 months of age, after which all visits will be relative to the patient's date of birth. Note: Depending on the patient's age at dosing, the duration of participation at the end-of-trial visit can vary from approximately 12 months (baby dosed at approximately 6 months of age) to approximately 18 months (baby dosed near birth "0 months of age").

Investigational Product: AVXS-101


following treatment guideline: taper from 1 mg/kg/day to 0.5 mg/kg/day during Weeks 5 and 6 post-AVXS-101 infusion, then taper to 0.25 mg/kg/day during Weeks 7 and 8, and then discontinue prednisolone at Week 9.

Efficacy will be assessed by achievement of the key developmental milestone of sitting without support for at least 10 seconds at any time up to and including the 18 month of age trial visit and survival at 14 months of age (as defined in Section 14.1.1.1.1). Safety will be assessed through monitoring AEs, concomitant medication usage, physical examinations, vital sign assessments, cardiac assessments, and laboratory evaluations (Section 12).

Additionally, a Data Safety Monitoring Board/Data Monitoring Committee (DSMB/DMC) will review safety data on a quarterly basis. A detailed description of the DSMB/DMC, its role in this trial, and the timing and process of the scheduled reviews will be described in a DSMB/DMC Charter.

# 7.2. Number of Patients

Thirty patients are planned to enroll. Patients who are in screening and meet eligibility criteria for the study when the enrollment target is met may be enrolled upon approval of the sponsor.

### 7.3. Criteria for Trial Termination

An independent DSMB/DMC will conduct quarterly and ad hoc reviews of the emerging safety data throughout the trial as described in Section 15.

The trial may be terminated for the following reasons:

- Development of unacceptable toxicity, defined as the occurrence of any unanticipated CTCAE Grade 3 or higher AE/toxicity that is possibly, probably, or definitely related to gene replacement therapy, and is associated with clinical symptoms and/or requires medical treatment.
- DSMB/DMC can recommend early termination of the trial for safety reasons.
- Trial is terminated by Sponsor.
- Regulatory Authority recommendation.


#### 8. SELECTION AND WITHDRAWAL OF PATIENTS

Patients with SMA Type 1 who are < 6 months (< 180 days) of age **at the time** of gene replacement therapy (Day 1) with proven biallelic mutations of the *SMN1* gene and 1 or 2 copies of the *SMN2* will be enrolled in this trial. Patients may be of any racial, ethnic, or gender background.

#### 8.1. Patient Inclusion Criteria

Patients must meet all of the following inclusion criteria:

- 1. Patients with SMA Type 1 as determined by diagnosis of SMA based on gene mutation analysis with biallelic SMN1 mutations (deletion or point mutations) and 1 or 2 copies of SMN2 [inclusive of the known SMN2 gene modifier mutation (c.859G>C)]
- 2. Patients must be < 6 months (< 180 days) of age at the time of AVXS-101 infusion
- 3. Patients must have a swallowing evaluation test performed prior to administration of gene replacement therapy
- 4. Up-to-date on childhood vaccinations that include palivizumab prophylaxis (also known as Synagis) to prevent RSV infections are also recommended.
- 5. Parent(s)/legal guardian(s) willing and able to complete the informed consent process and comply with trial procedures and visit schedule

#### 8.2. Patient Exclusion Criteria

Patients must not meet any of the following exclusion criteria:

- 1. Previous, planned or expected scoliosis repair surgery/procedure prior to 18 months of age
- 2. Use of invasive ventilatory support (tracheotomy with positive pressure) or pulse oximetry < 95% saturation at screening
  - a. Pulse oximetry saturation must not decrease ≥ 4 percentage points between screening and dosing with confirmatory oximetry reading
  - b. Patients may be put on non-invasive ventilatory support for < 12 hours per day at the discretion of their physician or trial staff
- 3. Use or requirement of non-invasive ventilatory support for ≥12 hours daily in the 2 weeks prior to dosing
- 4. Patient with signs of aspiration based on a swallowing test or whose weight-for-age falls below the 3<sup>rd</sup> percentile based on WHO Child Growth Standards [42] and unwilling to use an alternative method to oral feeding
- 5. Active viral infection (includes human immunodeficiency virus [HIV] or positive serology for hepatitis B or C, or known Zika virus infection)
- 6. Serious non-respiratory tract illness requiring systemic treatment and/or hospitalization within 2 weeks prior to screening

Investigational Product: AVXS-101


- 7. Upper or lower respiratory infection requiring medical attention, medical intervention, or increase in supportive care of any manner within 4 weeks prior to screening
- 8. Severe non-pulmonary/respiratory tract infection (e.g., pyelonephritis, or meningitis) within 4 weeks before administration of gene replacement therapy or concomitant illness that, in the opinion of the Principal Investigator, creates unnecessary risks for gene replacement such as:
  - a. Major renal or hepatic impairment
  - b. Known seizure disorder
  - c. Diabetes mellitus
  - d. Idiopathic hypocalcuria
  - e. Symptomatic cardiomyopathy
- 9. Known allergy or hypersensitivity to prednisolone or other glucocorticosteroids or their excipients.
- 10. Concomitant use of any of the following: drugs for treatment of myopathy or neuropathy, agents used to treat diabetes mellitus, or ongoing immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, or immunosuppressive therapy within 3 months prior to gene replacement therapy (e.g., corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, IV immunoglobulin, rituximab)
- 11. Anti-AAV9 antibody titer > 1:50 as determined by Enzyme-linked Immunosorbent Assay (ELISA) binding immunoassay. Should a potential patient demonstrate Anti-AAV9 antibody titer > 1:50, he or she may receive retesting within 30 days of the screening period and will be eligible to participate if the Anti-AAV9 antibody titer upon retesting is ≤ 1:50
- 12. Clinically significant abnormal laboratory values (GGT, ALT, and AST, or total bilirubin > 2 × ULN, creatinine ≥ 1.0 mg/dL, hemoglobin [Hgb] < 8 or > 18 g/dL; white blood cell > 20,000 per cmm) prior to gene replacement therapy. Patients with an elevated bilirubin level that is unequivocally the result of neonatal jaundice shall not be excluded.
- 13. Participation in recent SMA treatment clinical trial (with the exception of observational Cohort studies or non-interventional studies) or receipt of an investigational or commercial compound, product or therapy administered with the intent to treat SMA (e.g., nusinersen, valproic acid) at any time prior to screening for this trial. Oral beta-agonists must be discontinued at least 30 days prior to dosing. Inhaled albuterol specifically prescribed for the purposes of respiratory (bronchodilator) management is acceptable and not a contraindication at any time prior to screening for this trial.
- 14. Expectation of major surgical procedures during the trial assessment period (e.g., spinal surgery or tracheostomy)
- 15. Parent(s)/legal guardian(s) unable or unwilling to comply with trial procedures or inability to travel for repeat visits

Investigational Product: AVXS-101


- 16. Parent(s)/legal guardian(s) unwilling to keep trial results/observations confidential or to refrain from posting confidential trial results/observations on social media sites
- 17. Parent(s)/legal guardian(s) refuses to sign consent form
- 18. Patients < 35 weeks gestational age at time of birth

#### 8.3. Patient Withdrawal Criteria

Patients may be discontinued from the trial for the following reasons:

- Death
  - An autopsy and/or post-mortem tissue/organ collection will be requested for any patient who expires following participation (see Post-Mortem Tissue and Organ Collection Plan in Appendix 2)
- Failure to comply with protocol-required visits or trial procedures for 3 or more consecutive visits that are not rescheduled, unless due to hospitalization
- Parent(s)/legal guardian(s) withdraws consent
- Investigator discretion

End-of-Trial procedures should be completed within 14 days for any patient who prematurely discontinues the trial for any reason, as indicated in Appendix 1. Patients who terminate the study early for reasons other than death will be offered enrollment in a long-term follow-up study.

In instances in which a patient withdraws from the study prior to the last scheduled visit, the investigator should differentiate between factors that are related to a catastrophe (such as the inability to travel, local ordinances or other restrictions, etc.) versus withdrawal of consent.


# 9. TREATMENT OF PATIENTS

It is the responsibility of the Investigator to ensure the safe storage and administration of gene replacement therapy.

## 9.1. Description of Trial Product

AVXS-101 is a non-replicating recombinant AAV9 containing the *SMN* gene under the control of the cytomegalovirus (CMV) enhancer/ CB. One of the 2 AAV inverted terminal repeats (ITRs) has been modified to promote intramolecular annealing of the transgene, thus forming a double stranded transgene ready for transcription.

**Table 2: Investigational Product** 

| | Investigational Product |
|---|---|
| Product Name | AVXS-101 |
| Unit Dose | $1.1 \times 10^{14}$ vg/kg; Equivalent to the dose received by the Cohort 2 in the Phase 1 study (AVXS-101-CL-101) as determined by direct product testing with improved analytical methods. |
| Route of Administration | Intravenous infusion |
| Physical Description | AVXS-101 is a clear, colorless to faint white solution. |

#### 9.2. Prior and Concomitant Medications

Prior and concomitant medications will be captured in the electronic Case Report Form (eCRF) from 2 weeks prior to administration of gene replacement therapy through the last trial visit.

#### 9.2.1. Prophylactic Administration of Prednisolone

An antigen specific T-cell response to the AAV vector was observed in the completed Phase 1 clinical trial (AVXS-101-CL-101) investigating AVXS-101 treatment via IV infusion [data on file]. This is an expected response between 2 to 4 weeks following gene replacement therapy. One possible consequence to such antigen specific T-cell response is clearance of the transduced cells and loss of transgene expression.

In an attempt to dampen the host immune response to the AAV based therapy, all patients will receive prophylactic prednisolone at approximately 2 mg/kg/day (or an equivalent dose of another glucocorticoid if prednisolone is unavailable or in the opinion of the investigator prednisolone is not tolerated [41]) on Day -1, Day 1, and Day 2, and then 1 mg/kg/day starting on Day 3 and until at least 30 days post-AVXS-101 infusion. After 30 days post-AVXS-101 infusion, the dose of prednisolone can be tapered for patients whose GGT, ALT, and AST values are below the threshold of 2 × ULN. To summarize, the overall course of prednisolone should follow the following treatment guideline:

- Day -1, Day 1, and Day 2: 2 mg/kg/day
- Day 3 until at least 30 days post AVXS-101 infusion: 1 mg/kg/day


- Weeks 5 and 6 post-AVXS-101 infusion: 0.5 mg/kg/day
- Weeks 7 and 8 post-AVXS-101 infusion: 0.25 mg/kg/day
- Week 9 post-AVXS-101 infusion: prednisolone discontinued

Liver function testing should guide each step of the taper, and liver function tests should be checked prior to prednisolone discontinuation. If the GGT, AST, or ALT values are ≥2 × ULN, then the present dose of prednisolone will be adjusted as needed until the GGT, AST, and ALT values decrease below threshold, at which point the taper may continue. Liver function tests should also be checked approximately 2 weeks after the taper has concluded and prednisolone has been discontinued to evaluate for rebound elevation of GGT, AST, or ALT levels. Variance from these recommendations will be at the discretion of the Investigator based on potential safety issues for each patient. If another glucocorticoid is used in place of prednisolone by the Investigator, similar considerations should be taken into account after 30 days and tapered as appropriate and at the discretion of the Investigator.

#### 9.2.2. Prohibited Medications

Concomitant use of any of the following medications is prohibited:

- Drugs for treatment of myopathy or neuropathy, or agents used to treat diabetes mellitus
- Therapy received with the intent to treat SMA (e.g., nusinersen, valproic acid); oral β-agonists must be discontinued at least 30 days prior to gene therapy dosing. Inhaled β-agonists may be used to treat respiratory complications of SMA provided such medications are dosed at clinically appropriate levels
- Any investigational medication other than AVXS-101 is prohibited during the trial
- Ongoing immunosuppressive therapy, plasmapheresis, immunomodulators such as adalimumab, or immunosuppressive therapy within 3 months prior to AVXS-101 dosing (e.g., corticosteroids, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, IV immunoglobulin, rituximab)

Corticosteroid usage following completion of the prednisolone taper is permissible as part of routine clinical management. The use of corticosteroids in such circumstances should be documented appropriately as a concomitant medication, and the event precipitating its usage should be appropriately documented as an adverse event.

Should the use of corticosteroids (aside from inhaled corticosteroids for bronchospasm) be considered as part of care during the course of the prednisolone taper, this medical management should be discussed with the medical monitor.

#### 9.2.3. Vaccinations

Where feasible, the vaccination schedule should be adjusted appropriately to accommodate the prednisolone use. When avoiding vaccination while on steroids represents an undue delay or interruption of a vaccination schedule, vaccination should continue at the discretion and judgement of the treating physician given 1) the importance of maintaining childhood

Investigational Product: AVXS-101


vaccination in this population and 2) the published literature that indicates that vaccination while on steroid doses 1 mg/kg/day or below is safe and effective [43].

Vaccinations that include palivizumab (also known as Synagis®) prophylaxis to prevent respiratory syncytial virus infections are also recommended (31, 44).

## 9.3. Treatment Compliance

AVXS-101 will be administered as a one-time IV injection.

# 9.4. Randomization and Blinding

This is an open-label trial.


#### 10. TRIAL PRODUCT MATERIALS AND MANAGEMENT

AVXS-101 is manufactured in accordance with current Good Manufacturing Practices (cGMP).

## 10.1. Trial Product

AVXS-101

#### **10.2.** Trial Product Dose and Dose Justification

Patients will receive a 1-time dose of AVXS-101 at  $1.1 \times 10^{14}$  vg/kg, equivalent to the dose received by Cohort 2 in the Phase 1 study via IV infusion administered in the completed Phase 1 clinical study (AVXS-101-CL-101).

Two doses were studied in the completed Phase 1 clinical study (AVXS-101-CL-101); the higher dose (dose received by the Cohort 2 patients) was chosen for the present study as preliminary data demonstrated both a dose response and significant clinical benefit thus identifying it as the proposed therapeutic dose. In the Phase 1 study, AVXS-101 demonstrated a dose response, with efficacy greater as observed by motor milestone achievement and CHOP INTEND scores at the higher dose (received by Cohort 2) than at the lower dose (received by Cohort 1). Direct testing of the actual lot of Investigational Medicinal Product (IMP) used in the AVXS-101-CL-101 study by an improved and more fully qualified analytical method has assigned a value of  $1.1 \times 10^{14}$  vg/kg to the actual dose received by Cohort 2 in this Phase 1 study. The same method has been used to establish an equivalent dose for the Phase 3 IMP. This vg/kg value has been further verified in an improved and more fully qualified SMN $\Delta$ 7 Mouse Biopotency assay to support a similar extension of mouse lifetime in direct comparative assessment between the Phase 1 and Phase 3 IMP.

# 10.3. Trial Product Packaging and Labeling

AVXS-101 kits will be labeled with a specific kit number and batch/lot number assigned at the cGMP facility. The content of the labeling is in accordance with the local regulatory specifications and requirements.

# 10.4. Trial Product Storage and Destruction

AVXS-101 kits will be stored in a locked, limited access room under the responsibility of the Investigator or other authorized persons (e.g., pharmacists) in accordance with local regulations, policies, and procedures. Control of storage conditions, especially control of temperature (e.g., refrigerated/freezer storage) and information on in-use stability and instructions for handling prepared AVXS-101 should be managed in accordance with the Pharmacy Manual.

The vessel used for delivery of the vector should be resealed in the procedure room and processed for destruction in accordance with the Pharmacy Manual and applicable biohazardous waste guidelines for disposal.


# 10.5. Trial Product Preparation

Preparation of AVXS-101 will be done aseptically under sterile conditions and will be received ready for infusion.

AVXS-101 will arrive as outlined in the Pharmacy Manual. The total vector genome dose will be calculated based on the patient's body weight.

The dose-delivery vessel will be delivered to the designated pediatric intensive care unit (PICU), patient room or other appropriate setting (e.g., interventional suite, operating room, dedicated procedure room) with immediate access to acute critical care management. The vessel will be delivered in accordance with the Pharmacy Manual.

#### 10.6. Trial Product Administration

AVXS-101 infusion will be administered under sterile conditions in a PICU or other appropriate setting (e.g., interventional suite, operating room, dedicated procedure room) with immediate access to acute critical care management. AVXS-101 will be delivered 1-time through a venous catheter inserted into a peripheral limb vein (arm or leg) at a dose equivalent to the Cohort 2 dose administered in the AVXS-101-CL-101 trial. AVXS-101 should be slowly infused over approximately 60 minutes, dependent upon volume required, utilizing an infusion set and pump in accordance with the Pharmacy Manual.

Following administration of gene replacement therapy, patients should return to an appropriate designated setting to ensure close monitoring of vital signs and adverse events. Vital signs will be continuously monitored throughout the gene replacement therapy infusion as described in Section 12.1.3. Patients should be maintained in the PICU or other appropriate setting for 48 hours after the start of gene replacement therapy.

# 10.7. Dose Adjustment Criteria

The trial investigates a 1-time IV infusion of AVXS-101; no dose adjustments are possible.

# **10.8.** Trial Product Accountability

The pharmacist or designee will maintain accurate records of the quantities of AVXS-101 received, dispensed, destroyed, and/or returned to AveXis. The pharmacist or designee will document the date and time of delivery of the dose vessel to the dose procedure room as well as the time the used vessel was processed for destruction as per the Pharmacy Manual.

# 10.9. Trial Product Handling and Disposal

All materials used for injection, including sterile drapes, needles, and syringes in contact with the vector must be sealed in leak-proof containers. All waste must be sealed in bags bearing the biohazard symbol and disposed of in a biohazard waste container.

All transfers must be done in spill-proof containers. Individuals manipulating the vector will be required to wear personal protective equipment, such as gloves.

Investigational Product: AVXS-101


Any quality issue noticed with the receipt or use of AVXS-101 (e.g., deficiency in condition, appearance, pertaining to documentation, labeling, expiration date, etc.) should be promptly reported to the Sponsor in accordance with procedures outlined in the Pharmacy Manual.

Under no circumstances will the Investigator supply AVXS-101 to a third party, allow AVXS-101 to be used other than as directed by this clinical trial protocol, or dispose of AVXS-101 in any other manner.


#### 11. ASSESSMENT OF EFFICACY

Efficacy will be assessed by achievement of the key developmental milestone of sitting without support for at least 10 seconds at any time up to and including the 18 months of age trial visit and survival at 14 months of age (as defined in Section 14.1.1.1.1). Efficacy assessments will be performed at the times specified in the SoA (Appendix 1) and should be the first assessments performed at any scheduled visit. All post-treatment visits will be relative to the date on which gene replacement therapy is administered until the patient is 14 months of age after which all visits will be relative to the patient's date of birth.

In the event of unforeseen catastrophe or other, serious situation (such as the COVID-19 pandemic) that occurs during the study, which limits or prevents on-site study visits, alternative methods of data collection pertaining to efficacy assessments may be considered. Critical data that pertain to the coprimary and co-secondary endpoints should be collected according to the overall study schedule and within the protocol-defined visit window. The maintenance of the overall visit schedule and visit windows is especially important for the final scheduled study visit, as this may impact the overall interpretation of the evaluation of efficacy. As described in Section 7.1, allowances are made for the collection of data remotely, when necessary.

Video recordings demonstrating the attainment of any new developmental milestones should be obtained within the protocol-defined visit window, including those that are required to be assessed as part of the final study visit or are related to co-primary or co-secondary endpoints (e.g, sitting without support). This may include submission of recordings made by the family or others as described in Section 11.3.

Alternative methods of data collection for efficacy assessments depending on local regulations, institutional polices, and capabilities may include:

- developmental/motor efficacy assessments by a qualified clinical evaluator during a visit to the participant's home
- Home videos or other recordings which demonstrate the achievement of developmental milestones that are specified in the protocol, including those to be assessed at the final scheduled study visit
- use of ventilatory, cough or feeding support by the participant, evaluated during phone calls, virtual contacts (e.g. teleconsult) or visits by site staff/home nursing service to the participant's home, or during visits by the participant to a local hospital.

# 11.1. Developmental Milestones

Developmental milestones will be assessed according to the 6 gross motor milestones definitions from the World Health Organization Multicentre Growth Reference Study (WHO MGRS) (Appendix 5) [24] and the BSIDv03 and will be analyzed to assess efficacy (Appendix 3 and Appendix 4). Achievement of each developmental milestone will be determined by the qualified site clinical evaluator (physical or occupational therapist or national equivalent) and confirmed by the central reviewer based on an assessment of the submitted videotapes (Section 11.3). Developmental milestones will be determined at each visit as shown in the SoA (Appendix 1) and as described in Section 11.2.

Investigational Product: AVXS-101


At the 18 months of age visit all developmental milestones (Appendix 4 and Appendix 5) should be assessed, documented, and video recorded, regardless of previous attainment.

#### 11.2. Motor Function Tests

### 11.2.1. World Health Organization Multicentre Growth Reference Milestones

The World Health Organization Multicentre Growth Reference Trial Group milestones defined for this study include 6 gross motor milestones (Appendix 5):

- Sitting without support for 10 seconds, does not use arms or hands
- Crawling on hands and knees, at least 3 consecutive movements
- Standing with assistance at least 10 seconds
- Walking with assistance at least 5 steps
- Standing alone at least 10 seconds
- Walking alone at least 5 steps

These 6 gross milestones will be assessed by a qualified clinical evaluator according to the SoA (Appendix 1). If the Bayley Gross Motor Subtest Item 22 (Appendix 3), sits without support for 5 seconds, is achieved at a visit, then the WHO milestone for sitting without support for at least 10 seconds (Appendix 5) should be assessed at that visit and all subsequent visits. Each developmental milestone assessment will be evaluated according to the WHO defined performance criteria and will be video recorded in accordance with the AVXS-101-CL-302 Physical Assessments Manual and may be submitted for review by a central reader (Section 11.3).

### 11.2.2. Bayley Scales for Infant and Toddler Development/Developmental Milestones

The BSIDv03 (Appendix 3) is a standardized, norm-referenced infant assessment of developmental functioning across 5 domains of cognitive, language, motor, social-emotional, and adaptive behavior. The Bayley Scales will be administered by a qualified clinical evaluator in accordance with the Physical Assessments Manual. The items from BSIDv03 Gross Motor Subtest defined as developmental milestones for this protocol are specified in Appendix 4.

During the Screening visit, the clinical evaluator will complete an assessment of baseline developmental milestone achievement in accordance with Appendix 3; this assessment must address all developmental milestones/items noted in Appendix 3, Gross Motor Subtest that are at or below the child's baseline function, and be recorded on video. The findings must be documented in the source. Items that are below the baseline level of assessment that are not successfully achieved during the baseline evaluation should be repeated at subsequent visits until successfully performed.

The developmental milestone of functional independent sitting is defined by BSID GM#26, sitting for at least 30 seconds without external support from another person or object, however the child is allowed to use their upper extremities. This developmental milestone should be assessed, documented, and video recorded at every subsequent visit until attainment,

Investigational Product: AVXS-101


regardless of starting point on the scale. It must be assessed at the 18 months of age visit regardless of previous attainment.

The gross and fine motor subtests of the motor domain will be administered according to the SoA (Appendix 1).

Each Bayley Scales assessment will be video recorded in accordance with the AVXS-101-CL-302 Physical Assessments Manual, and videos containing developmental milestone evidence will be submitted for review by an independent central reviewer (Section 11.3).

#### 11.2.3. CHOP INTEND

The CHOP INTEND is a motor function scale developed and validated for use specifically to monitor motor function status and decline amongst children with SMA Type 1, and will be administered by a qualified clinical evaluator [45, 46]. The CHOP INTEND scale (Appendix 6) examines several aspects of motor function, including head control, righting reactions, and trunk movements in supported sitting, supine, and prone positions. Anti-gravity movements in assisted rolling, ventral suspension, and supported standing will also be measured. Additional information on contractures will also be collected as described in the Physical Assessments Manual.

The CHOP INTEND will be performed according to the SoA (Appendix 1). For purposes of efficacy assessments, the CHOP INTEND assessment performed at Day -1 will be treated as the baseline assessment.

Patients who achieve 3 consecutive CHOP INTEND scores  $\geq$  58 will not undergo any additional CHOP INTEND examinations.

Each CHOP INTEND exam will be video recorded in accordance with the AVXS-101-CL-302 Physical Assessments Manual (Section 11.3).

#### 11.3. Video Evidence

Clinic assessments (WHO Motor Developmental Milestones, Bayley Scales and CHOP INTEND) required at each trial visit will be video recorded in an effort to produce compelling, demonstrable, documented evidence of efficacy, as determined by changes in functional abilities. AveXis, Inc. (AveXis) will provide a secure and confidential upload process for transfer and storage of the videos from investigational sites to a contracted third-party vendor that will compile and arrange videos as per AveXis requirements. Any/all videos received at AveXis or the contracted vendor will be treated as confidential trial data and will be the sole property of AveXis. AveXis and the contracted vendor will provide this secure, encrypted transfer and storage solution to properly protect the identities of patients/families on the videos, which may be shared with regulatory agencies, the medical community, and/or in appropriate venues to discuss the results of this clinical trial.

All videos of Developmental Milestones which meet WHO and BSID criteria will be provided to an independent, central reviewer for unbiased assessment of developmental milestone achievement. The independent central reviewer will document whether the video displays

Investigational Product: AVXS-101


evidence of having achieved each developmental milestone. The date of developmental milestone achievement will be computed as the earliest date on which video evidence demonstrates the achievement of the specified developmental milestone.

At the 18 month of age visit, the WHO Motor Developmental Milestone for sitting without support for at least 10 seconds (Appendix 5) and BSID GM #26 – Sits without support for 30 seconds (Appendix 4) (functional independent sitting) will be submitted for central review, even if previously confirmed.

New developmental milestones attained for the first time at 18 months of age will also be submitted for central review.

Additionally, the parent(s)/legal guardian(s) may submit additional videos demonstrating achievement of developmental milestones at any time during the trial. These videos will be handled in the same manner in which the trial-derived videos are handled.


#### 12. ASSESSMENT OF SAFETY

In the event of unforeseen catastrophe or other, serious situation (such as the COVID-19 pandemic) that occurs during the study, which limits or prevents on-site study visits, regular phone or virtual video calls may occur (as per the Schedule of Assessments, every month or more frequently if needed) for safety monitoring and discussion of the participant's health status. Visits by site staff/home nursing service to the participant's home, or visits by the participant to a local hospital, laboratory, or imaging center, for performing certain safety assessments, depending on local regulations and capabilities, can replace on-site study visits, if necessary. Analysis of laboratory samples (e.g. chemistry, hematology, urinalysis) may be performed at a local laboratory, if it is not possible to follow the central laboratory process. Other safety assessments that cannot be conducted by telephone (such as vital signs, weight, length, cardiac testing etc.) may similarly be collected by the methods described above.

# 12.1. Safety Parameters

Safety parameters include physical examinations, pulmonary examinations, vital signs, capillary blood gas assessments, weight and length measurements, 12-lead ECGs, echocardiograms, 24-hour Holter monitors, swallowing tests, laboratory assessments, adverse event monitoring, and photographs of the infusion site. In general, safety assessments will be performed at the times specified in the SoA (Appendix 1). All post-treatment visits are relative to the date on which gene replacement therapy is administered until the patient is 14 months of age, after which all visits will be relative to the patient's date of birth.

# 12.1.1. Demographic/Medical History

Demographic/medical history information will be collected at screening and captured in the eCRF. Information that will be collected includes:

- Familial history of SMA including affected siblings or parent carriers
- Gestational age at birth
- Length/height/head circumference at birth
- Hospitalization information from time of birth including number, duration, and reason for hospitalizations including International Statistical Classification of Diseases and Related Health Problems (ICD-10 codes), if available
- Historical ventilator support, if any
- Historical feeding support, if any.

Patients are encouraged to follow all routinely scheduled immunizations, as recommended by the Local European Guideline throughout the trial. Vaccinations that include palivizumab prophylaxis (also known as Synagis) to prevent RSV infections are also recommended.

#### 12.1.2. Physical Examinations

Physical examinations will be conducted by the Investigator or designee as specified in the SoA (Appendix 1). The Day 1 physical examination will be performed prior to the start of gene replacement therapy infusion. Physical examinations include a review of the following systems:

Investigational Product: AVXS-101


head, eyes, ears, nose and throat (HEENT), lungs/thorax, cardiovascular, abdomen, musculoskeletal, dermatologic, lymphatic, neurologic, and genitourinary. Specifically, the neurological exam should include detailed, age-appropriate sensory testing (such as examination of proprioceptive, vibratory, tactile and pain sensation) at each visit. Any clinically significant abnormal finding should be recorded as an adverse event. Further clinical evaluation should be considered per judgment of the investigator.

The head circumference shall be measured with each physical examination. To measure head circumference, the examiner should securely wrap a flexible measuring tape around the circumference of the head, above the eyebrows over the broadest part of the forehead, above the ears, and over the most prominent part of the occiput. The measurement should be taken 3 times, and the largest measurement should be recorded to an accuracy of 0.1 centimeters.

#### 12.1.3. Vital Signs/Weight and Length

Vital sign parameters include blood pressure, respiratory rate, pulse, temperature, and pulse oximetry. Vital signs will be obtained as specified in the SoA (Appendix 1). On Day 1, vital signs will be continuously monitored throughout the gene replacement therapy infusion and recorded pre-dose and every 15 ( $\pm$  5) minutes from the start of the infusion for the first 4 hours after the start of infusion, and then every hour ( $\pm$  15 minutes) until 24 hours after the start of infusion. Temperature will be recorded pre- and post-infusion.

Weight and length will be measured at each trial visit as specified in the SoA (Appendix 1). On Day 1, weight and length will be measured pre-dose.

#### 12.1.4. Electrocardiogram

A 12-lead ECG will be performed as specified in the SoA (Appendix 1).

For patients who were previously following the 6-monthly ECG schedule, a 12-lead ECG is to be performed at the study visit during which consent for additional ECGs is first obtained (ICF corresponding to protocol version 3.0 or later) and then in accordance with the SoA. Additional electrophysiological monitoring will be at the discretion of the Investigator as per local institutional guidelines

The ECG will be interpreted locally by a cardiologist or designee for immediate safety evaluation. The ECG tracings or ECG machine data will also be collected for centralized review and interpretation by a cardiologist.

#### 12.1.5. Echocardiogram

A standard transthoracic echocardiogram will be performed as specified in the SoA (Appendix 1).

For patients who were previously following the 6-monthly echocardiogram schedule, an echocardiogram is to be performed at the study visit during which consent for additional echocardiograms is first obtained (ICF corresponding to protocol version 3.0 or later) and then in accordance with the SoA (Appendix 1).

Investigational Product: AVXS-101


The echocardiogram will be interpreted locally by a cardiologist or designee for immediate safety evaluation. The echocardiograms will also be collected for centralized review and interpretation by a cardiologist.

## 12.1.6. Continuous ECG Recordings

Twenty-four (24)-hour Holter monitoring will take place as specified in the SoA (Appendix 1).

For patients not already undergoing Holter monitoring from 3 months of age, 24-hour Holter monitoring will be performed when consent for additional recording is first obtained (ICF corresponding to protocol version 3.0 or later version).

Holter monitors will be provided to study sites along with a dedicated laptop for uploading the data from the memory cards for centralized review and analysis by a cardiologist or designee within 24 hours of data upload. AveXis will be notified of any safety concerns from the centralized review (Appendix 1).

## 12.1.7. Pulmonary Examinations

Pulmonary examinations will be performed by a pulmonologist (or appropriate individual as per standard institutional practice) as specified in the SoA (Appendix 1). Prior to trial entry, a pulmonologist (or appropriate individual as per standard institutional practice) will review and document ventilator usage in the 2 weeks prior to screening.

Patients may be fitted with non-invasive ventilator support at the discretion of the pulmonologist (or appropriate individual as per standard institutional practice) and/or Investigator. Non-invasive ventilator support equipment will be provided by AveXis, Inc. through a third-party vendor if not covered by the patient's insurance.

Should the patient require non-invasive ventilator support at any time during the trial, the usage should be recorded in eCRF. Patients requiring non-invasive ventilator support will be asked to bring the machine to each trial visit.

#### 12.1.8. Swallowing Test

A standard bedside, non-barium (unless required per institutional policy), swallowing test will be performed as specified in the SoA (Appendix 1) to determine if the patient has signs of aspiration. The swallowing test at Screening can be performed at the investigator site. If the test is positive for aspiration, there may be a recommendation for the patient to use an alternate method to oral feeding for the duration of the trial at the determination of the Investigator and treating clinician.

#### 12.1.9. Photographs of Infusion Site

Photographs will be taken of the infusion site as specified in the SoA (Appendix 1) to monitor healing of the infusion site. The Day 1 infusion site photograph will be performed prior to the start of gene replacement therapy infusion. AveXis will provide a secure and confidential upload process for transfer and storage of the photographs from the investigative sites to a contracted third-party vendor that will compile and arrange photographs as per AveXis requirements. Any/all photographs received at AveXis or the contracted vendor will be treated as confidential

Investigational Product: AVXS-101


trial data and will be the sole property of AveXis. AveXis and the contracted vendor will provide this secure, encrypted transfer and storage solution to properly protect the identities of patients/families in the photographs, which may be shared with regulatory agencies, the medical community, and/or in appropriate venues to discuss the results of this clinical trial.

#### 12.1.10. Laboratory Assessments

Blood samples will be collected at each scheduled visit as specified in the SoA (Appendix 1) and in according with laboratory manuals provided for this study. On Day -1, required blood samples will be collected locally prior to the start of gene replacement therapy infusion; duplicate samples will not be collected for shipment to the central laboratory. Any clinically significant laboratory value will be repeated at the discretion of the Investigator.

In most instances, blood samples will be collected and shipped to a central laboratory; however, at the discretion of the Investigator, samples may be processed locally for emergent safety monitoring or other logistical or technical reasons that warrant samples to be processed locally. Samples for laboratory tests required during the in-patient AVXS-101 infusion period prior to dosing will be collected and processed by the investigative site's local laboratory to ensure receipt of results prior to dosing.

**Table 3: Total Blood Volume** 

| Visit | Tests <sup>a</sup> | Total Volume (mL) <sup>b</sup> |
|---|---|---|
| Screening | Hematology, chemistry/CK-MB or Troponin I, virus serology, ELISA immunology sample (AAV9/SMN Ab only), diagnostic genetic re-confirmation sample | 15.4 |
| Day 1 | Hematology, chemistry, capillary blood gas | 3.3 |
| Day 2 | Hematology, chemistry, capillary blood gas | 3.3 |
| Day 7 | Hematology, chemistry/CK-MB or Troponin I, immunology sample (ELISA) | 9.6 |
| Day 14 | Hematology, chemistry, immunology sample (ELISA only) | 3.3 |
| Day 21 | Hematology, chemistry, immunology sample (ELISA only) | 3.3 |
| Day 30 | Hematology, chemistry/CK-MB or Troponin I, immunology sample (ELISA) | 9.6 |
| Day 44 | Chemistry | 1.3ª |
| Day 60 | Hematology, Chemistry/CK-MB or Troponin I | 3.6 |
| Day 72 | Chemistry | 1.3 |
| Month 3/4/5/7/8/<br>10/11/13/14/16/1<br>7 | Hematology, chemistry | 26.6 |
| Month 6/9/12/15 | Hematology, chemistry/CK-MB or Troponin I | 14.4 |
| End of Trial/ET | Hematology, chemistry/CK-MB or Troponin I | 3.6 |

Investigational Product: AVXS-101


| Visit | Tests <sup>a</sup> | Total Volume (mL) <sup>b</sup> |
|---|---|---|
| Maximum Total Volume for Trial <sup>c</sup> | | 98.6 |

CK-MB = creatinine kinase-muscle/brain; ET = early termination

In a case where sufficient blood cannot be collected from a patient, blood will be used in the following priority order with the first having greatest priority and last having the least priority:

- 1. Safety labs: chemistry → hematology → creatinine kinase-muscle/brain (CK-MB) or Troponin I
- 2. Serum antibody to AAV9 and SMN
- 3. Genetic reconfirmation testing

If there is insufficient blood volume to include the genetic reconfirmation testing sample at the screening visit, patient must return before Visit 2. All patients must have genetic reconfirmation testing completed.

#### **12.1.10.1.** Hematology

Hematology analysis will include a complete blood count with differential and platelet count with smear. Samples will be collected and shipped in accordance with the laboratory manual provided by the central laboratory. Blood samples for hematology analysis will be collected as specified in the SoA (Appendix 1).

Immediate/same-day hematology analyses required during in-patient dosing, as determined by Investigator, will be performed as per investigational site standard procedures at the local laboratory. Investigators will receive hematology results from all trial visits from the central laboratory.

### 12.1.10.2. Blood Chemistry

Samples will be collected and shipped in accordance with the laboratory manual provided by the central laboratory. Blood samples for chemistry analysis will be collected as specified in the SoA (Appendix 1).

Immediate/same-day chemistry analyses required during in-patient dosing, as determined by Investigator, will be performed as per investigational site standard procedures at the local laboratory.

Chemistry analysis will include the following at all trial visits:

<sup>&</sup>lt;sup>a</sup> Patients screened and dosed before IRB/EC approval of Protocol version 3.0 incorporating Amendment 2 will be tested for CK-MB throughout the study. Patients screened before IRB/EC approval of Protocol version 3.0 incorporating Amendment 2 but dosed afterwards will be tested for CK-MB at screening but for Troponin 1 at baseline and thereafter. Patients screened after IRB/EC approval of Protocol version 3.0 incorporating Amendment 2 will be tested for Troponin 1 from screening onwards.

<sup>&</sup>lt;sup>b</sup> Troponin I requires 0.3 mL less blood than CK-MB, thus total blood volumes will be less for participants receiving troponin I testing.

<sup>&</sup>lt;sup>c</sup> Patients will have different numbers of monthly visits, depending on their age at dosing. Maximum total volume based on a maximum of 16 monthly visits. Additionally, lower blood volumes may be sufficient at some visits where testing can be combined.

Investigational Product: AVXS-101


- Serum GGT
- AST/ALT
- Serum total bilirubin
- Direct bilirubin
- Albumin
- Glucose
- Creatinine kinase
- Creatinine
- BUN
- Electrolytes
- Alkaline phosphatase

CK-MB or Troponin I will be collected as specified in the SoA (Appendix 1) as applicable:

- Patients screened and dosed before IRB/EC approval of Protocol version 3.0 incorporating Amendment 2 will be tested for CK-MB throughout the study.
- Patients screened before IRB/EC approval of Protocol version 3.0 incorporating Amendment 2 but dosed afterwards will be tested for CK-MB at screening but for Troponin 1 at baseline and thereafter.
- Patients screened after IRB/EC approval of Protocol version 3.0 incorporating Amendment 2 will be tested for Troponin 1 from screening onwards.

Investigators will receive chemistry results from all trial visits from the central laboratory.

#### 12.1.10.3. Urinalysis

Urine samples will be collected in accordance with the laboratory manual provided by the central laboratory as specified in the SoA (Appendix 1). Day -1 urinalysis will be processed locally in accord with local procedures. Urinalysis will include the following parameters:

- Color
- Clarity/turbidity
- pH
- Specific gravity
- Glucose
- Ketones
- Nitrites
- Leukocyte esterase

Investigational Product: AVXS-101


- Bilirubin
- Blood
- Protein
- Red Blood Cell
- White Blood Cell
- Squamous epithelial cells
- Casts
- Crystals
- Bacteria
- Yeast

## 12.1.10.4. Virus Serology

The administration of an AAV vector has the risk of causing immune-mediated hepatitis. For patients who have HIV or positive serology for hepatitis B or C, administration of AAV vector may represent an unreasonable risk; therefore, negative serology testing must be confirmed at screening, prior to treatment. These samples will be collected at screening (Appendix 1) and shipped in accordance with the laboratory manual provided by the central laboratory.

# 12.1.10.5. Capillary Blood Gas

Capillary blood gas will be completed locally at Day –1 and Day 2 (Appendix 1). A puncture or small incision will be made with a lancet or similar device into the cutaneous layer of the patient's skin at a highly vascularized area (heel, finger, toe). To accelerate blood flow and reduce the difference between the arterial and venous gas pressures, the area will be warmed prior to the puncture. As the blood flows freely from the puncture site, the sample will be collected in a capillary tube.

#### 12.1.10.6. Immunology Testing (ELISA)

Blood samples for immunology testing will be collected and shipped to the central laboratory in accordance with the laboratory manual to test for serum antibodies to AAV9 and SMN (ELISA). Blood samples will be collected as specified in the SoA (Appendix 1).

#### 12.1.10.7. AAV9 Antibody Screen in Biological Mother

There is potential that the biological mother of the patient may have pre-existing antibodies to AAV9 that may be transferred to the patient through breast milk or, theoretically, via placental transfer in utero. Informed consent will be requested from the biological mother of the patient to screen the biological mother for circulating antibodies to AAV9. Once informed consent has been obtained, the biological mother will have her blood drawn from a peripheral vein at screening and shipped to the central laboratory for screening of anti-AAV9 antibodies. Patients whose biological mothers are involved with their care but do not consent to AAV9 antibody screening are not eligible to participate.

Investigational Product: AVXS-101


If AAV9 antibodies are identified, the Investigator should discuss with the biological mother whether to continue or to stop breast feeding. Patients consuming banked breast milk from donor sources that cannot be test for anti-AAV9 antibodies must be transitioned to formula prior to participation.

### 12.1.10.8. Blood for Diagnostic Confirmation Testing

A blood sample will be collected during the screening visit and shipped to the central laboratory in accordance with the laboratory manual for reconfirmation of *SMN1* deletions/mutations, *SMN2* copy number, and absence or presence of exon 7 gene modifier mutation (c.859G>C).

This will be done to ensure consistency in diagnostic testing practices.

#### 12.1.10.9. Saliva, Urine, and Stool Collection

Studies have shown that some vector can be excreted from the body for a few weeks after injection; this is called "viral shedding." Vector shedding can be found in the blood, urine, saliva, and stool for up to a few weeks following infusion. The risks associated with the shed vector are not known at this time; however, the risk is thought to be low as the vector cannot replicate. Regardless, IRB/IEC- approved instructions should be provided to the patient's family and care giver(s) regarding use of protective gloves if/when they come into direct contact with the patient's bodily fluids and/or waste, as well as good hand-hygiene for a minimum of 4 weeks after gene replacement therapy. Additionally, patients are prohibited from donating blood for 2 years following the vector infusion.

Saliva, urine, and stool samples will be collected for viral shedding studies as specified in the SoA (Appendix 1). Samples will be collected, prepared, and shipped as per the laboratory manual.


#### 13. ADVERSE AND SERIOUS ADVERSE EVENTS

## 13.1. Definition of Adverse Events

#### 13.1.1. Adverse Event

An AE is the development of an undesirable medical condition or the deterioration of a preexisting medical condition following or during exposure to a pharmaceutical product, whether or not considered casually related to the product. In clinical studies, an AE can include an undesirable medical condition occurring at any time, including baseline or washout periods, even if no trial treatment has been administered.

All AEs (related or not related) that occur after signing of the informed consent through the last trial visit will be collected and recorded in the eCRF.

All AEs will be classified in accordance with the CTCAE version 4.03 outlined in Table 4.

**Table 4: Common Terminology Criteria for Adverse Events** 

| Grade | Definition |
|---|---|
| 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental |
| | ADL. <sup>a</sup> |
| 3 | Severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of |
| | hospitalization indicated; disabling; limiting self-care ADL.b |
| 4 | Life-threatening consequences; urgent intervention indicated. |
| 5 | Death related to AE. |

Source: Common Terminology Criteria for Adverse Events (version 4.03) [40]

Additionally, a DSMB/DMC will review safety data on a quarterly basis. A detailed description of the DSMB/DMC, its role in this trial, and the timing and process of the scheduled reviews will be described in a DSMB/DMC Charter.

#### 13.1.2. Serious Adverse Event

A serious adverse event (SAE) is an AE occurring during any trial Phase (i.e., baseline, treatment, washout, or follow-up), and at any dose of the investigational product, or comparator that fulfils  $\geq 1$  of the following:

- Results in death
- It is immediately life-threatening
- It requires in-patient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability or incapacity

Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

b Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

Investigational Product: AVXS-101


- Results in a congenital abnormality or birth defect
- It is an important medical event that may jeopardize the patient or may require medical intervention to prevent one of the outcomes listed above.

All SAEs (related and not related) that occur after signing of the informed consent through 30 days after the last trial visit will be collected and recorded on forms provided by AveXis within 24 hours of the site becoming aware.

### 13.1.3. Adverse Events of Special Interest

The following are considered AEs of special interest (AESIs):

- Hepatotoxicity
- Thrombocytopenia
- Cardiac adverse events
- Sensory abnormalities suggestive of ganglionopathy

All AESIs (related and not related) that occur after signing of the informed consent through 30 days after the last study visit, irrespective of grade, should be collected and recorded on forms provided by AveXis within 24 hours of the site becoming aware.

# 13.2. Relationship to Trial Drug

An Investigator who is qualified in medicine must make the determination of relationship to the investigational product for each AE (Unrelated, Possibly Related, Probably Related, or Definitely Related). The Investigator should decide whether, in his or her medical judgment, there is a reasonable possibility that the event may have been caused by the investigational product. If no valid reason exists for suggesting a relationship, then the AE should be classified as "unrelated." If there is any valid reason, even if undetermined, for suspecting a possible cause-and-effect relationship between the investigational product and the occurrence of the AE, then the AE should be considered "related."

If the relationship between the AE/SAE and the investigational product is determined to be "possible" or "probable" then the event will be considered related to the investigational product for the purposes of expedited regulatory reporting.

# 13.3. Recording Adverse Events

Adverse events spontaneously reported by the patient and/or in response to an open question from the trial personnel or revealed by observation will be recorded during the trial at the investigational site. Information about AEs (related and not related) after signing of the informed consent form through the last study visit are to be collected. Serious adverse event information will be collected after signing of the informed consent form through 30 days after the last study visit. The AE term should be reported in standard medical terminology when possible. For each AE, the Investigator will evaluate and report the onset (date and time [if start date during inpatient period]), resolution (date and time [if start date during inpatient period]),

Investigational Product: AVXS-101


intensity, causality, action taken, serious outcome (if applicable), and whether or not it caused the patient to discontinue the trial.

It is important to distinguish between serious and severe AEs. Severity is a measure of intensity whereas seriousness is defined by the criteria under Section 13.1.2. An AE of severe intensity may not be considered serious.

## 13.4. Reporting Adverse Events

All SAEs (related and unrelated) will be recorded from signing of consent form through 30 days after the last trial visit. Any SAEs considered possibly, probably, or definitely related to the investigational product and discovered by the Investigator at any time after the trial should be reported. All SAEs must be reported to AveXis or designee within 24 hours of the first awareness of the event. The Investigator must complete, sign and date the SAE pages, verify the accuracy of the information recorded on the SAE pages with the corresponding source documents, and send a copy by fax or e-mail to AveXis or designee. Note: elective procedures or minor surgeries where hospitalization is required should not be reported as SAEs.

Additional follow-up information, if required or available, should all be faxed or e-mailed to AveXis or designee within 24 hours of receipt and this should be completed on a follow-up SAE form and placed with the original SAE information and kept with the appropriate section of the eCRF and/or trial file.

AveXis is responsible for notifying the relevant regulatory authorities of certain events. It is the Principal Investigator's responsibility to notify the IRB/IEC of all SAEs that occur at his or her site. Investigators will also be notified of all unexpected, serious, drug-related events (7/15 Day Safety Reports) that occur during the clinical trial. Each site is responsible for notifying its IRB/IEC of these additional SAEs.

# 13.5. Expedited Safety Reporting to Regulatory Authorities

All suspected, unexpected serious adverse reactions (SUSARs) will be reported to regulatory authorities within the 15—day expedited timeline. Fatal/life-threatening SUSARS will be reported immediately to French authorities and within the 7—day timeline to Eudravigilance according to EU regulation.


#### 14. STATISTICS

This section summarizes key aspects of the analysis plan including definitions of primary, secondary, and exploratory efficacy endpoints and safety endpoints, and the methods to be used to test the primary effectiveness hypothesis. Additional details regarding methods for the final data analysis will be provided in a separate Statistical Analysis Plan (SAP). The SAP will detail all analyses and data displays and will be executed according to Standard Operating Procedures in a controlled environment.

## 14.1. Data Analysis

#### 14.1.1. Trial Endpoints and Populations

#### 14.1.1.1. Trial Endpoints

The primary efficacy endpoint will be compared to the null. The secondary efficacy variable will be evaluated relative to literature-based historical controls (such as the PNCR) [24]. This variable was selected on the basis of comparability to the target population and similarity to the investigational device.

### 14.1.1.1. Primary Efficacy Endpoint

The primary efficacy endpoint is:

Proportion of symptomatic SMA Type 1 patients who are homozygous negative for *SMN1* exon 7 and have 2 copies of *SMN2* without the *SMN2* genetic modifier that achieve the ability to sit without support for at least 10 seconds at any visit up to and including the 18 months of age visit. It is defined by the WHO MGRS, confirmed by video recording, as a patient who sits up straight with head erect for at least 10 seconds; child does not use arms or hands to balance body or support position.

### 14.1.1.1.2. Secondary Efficacy Endpoint

The secondary efficacy endpoint is:

Survival at 14 months of age amongst symptomatic SMA Type 1 patients who are homozygous negative for *SMN1* exon 7 and have 2 copies of *SMN2* without the *SMN2* genetic modifier.

Survival is defined by the avoidance of the combined endpoint of either (a) death or (b) permanent ventilation, which is defined by tracheostomy or by the requirement of  $\geq$  16 hours of respiratory assistance per day (via non-invasive ventilator support) for  $\geq$  14 consecutive days in the absence of an acute reversible illness, excluding perioperative ventilation. Permanent ventilation, so defined, is considered a surrogate for death.

• An "acute reversible illness" is defined as any condition other than SMA that results in increased medical intervention (i.e., increased requirement for respiratory support; use of other concomitant medications as rescue) requirements and is expected to be reversible or improved following definitive intervention (i.e., surgery, antibiotics) or introduction of escalated supportive care, such as hospitalization (i.e., for upper respiratory infection, spontaneous fracture). The specific duration of the condition antecedent intervention

Investigational Product: AVXS-101


shall not be considered in the definition of "acute." The date of "definitive intervention" shall be defined as the date of provision of a procedure (i.e., surgery, etc.) or medication (i.e., antibiotics) intended to cure or substantially improve the condition. For conditions such as viral respiratory infections for which supportive care is provided, the date of "definitive intervention" shall be considered the date of hospitalization or substantial escalation of care.

- "Perioperative" use reflects any alteration of ventilator use related to a surgical or other medical procedure of any nature for which the patient received medications that could impair or interfere with respiratory function.
- For a patient who develops an acute reversible illness and/or requires perioperative ventilator support, a recovery period not to exceed 21 days following the date of definitive intervention will be instituted. Following this recovery period, the condition will be considered subacute and the patient will become evaluable with regards to the surrogate survival endpoint (requirement of ventilator support of ≥ 16 hours/day for 14 or more days).

### 14.1.1.1.3. Exploratory Endpoints

For the following exploratory efficacy endpoints, a Responder will be defined as a patient who demonstrates achievement of the endpoint at any post-procedure visit up to and including the 18-month trial visit.

- 1. Proportion of patients that achieve the ability to hold head erect without support as defined by BSIDv03 Gross Motor Subtest Item #4 (Appendix 3 and Appendix 4) [39].
- 2. Proportion of patients that achieve the ability to roll over as defined by BSIDv03 Gross Motor Subtest Item #20 (Appendix 3 and Appendix 4) [39].
- 3. Proportion of patients that achieve functional independent sitting for at least 30 seconds as defined by BSIDv03 Gross Motor Subtest Item #26, (Appendix 3 and Appendix 4) [39].
- 4. Proportion of patients that achieve the ability to stand with assistance for at least 2 seconds as defined by BSIDv03 Gross Motor Subtest Item #33 (Appendix 3 and Appendix 4) [39].
- 5. Proportion of patients that achieve the ability to crawl forwards on hands and knees for a distance of at least 5 feet as defined by BSIDv03 Gross Motor Subtest Item #34 (Appendix 3 and Appendix 4) [39].
- 6. Proportion of patients that achieve the ability to pull to standing as defined by BSIDv03 Gross Motor Subtest Item #35 (Appendix 3 and Appendix 4) [39].
- 7. Proportion of patients that achieve the ability to walk with assistance as defined by BSIDv03 Gross Motor Subtest Item #37 (Appendix 3 and Appendix 4) [39].
- 8. Proportion of patients that achieve the ability to stand alone for at least 3 seconds as defined by BSIDv03 Gross Motor Subtest Item #40 (Appendix 3 and Appendix 4) [39].
- 9. Proportion of patients that achieve the ability to walk at least 3 steps without support as defined by BSIDv03 Gross Motor Subtest Item #42 (Appendix 3 and Appendix 4) [39].

Investigational Product: AVXS-101


- 10. Proportion of patients that achieve the ability to crawl as defined by WHO Motor Developmental Milestones (Appendix 5) [38].
- 11. Proportion of patients that achieve the ability to stand with assistance as defined by WHO Motor Developmental Milestones (Appendix 5) [38].
- 12. Proportion of patients that achieve the ability to stand alone as defined by WHO Motor Developmental Milestones (Appendix 5) [38].
- 13. Proportion of patients that achieve the ability to walk with assistance as defined by WHO Motor Developmental Milestones (Appendix 5) [38].
- 14. Proportion of patients that achieve the ability to walk alone as defined by WHO Motor Developmental Milestones (Appendix 5) [38].
- 15. Improvement of raw score from baseline to the maximum using BSIDv03, Fine and Gross Motor Function Subtests (Appendix 3).
- 16. Maximum change from baseline in CHOP INTEND score (Appendix 6).
  - a. Proportion of patients achieving CHOP INTEND score  $\geq$  40 (Appendix 6).
  - b. Proportion of patients achieving CHOP INTEND score  $\geq$  50 (Appendix 6).
  - c. Proportion of patients achieving CHOP INTEND score  $\geq$  58 (Appendix 6).
- 17. Proportion of patients with the ability to remain independent of ventilator support, defined as requiring no daily ventilator support/usage at 18 months of age.
- 18. Proportion of patients maintaining the ability to swallow and to maintain weight (> third percentile based on WHO Child Growth Standards for age and gender [42]) without need of gastrostomy or other mechanical or non-oral nutritional support
- 19. Age at which patient first achieves WHO MGRS sitting without support (10 seconds) (Appendix 5)

### 14.1.1.1.4. Safety Endpoints

Assessment of the safety and tolerability of AVXS-101 treatment, including evaluation of AEs, laboratory data, vital signs, and concomitant medications.

#### 14.1.1.2. Statistical Analysis Populations

#### 14.1.1.2.1. Intent-to-Treat Population

The ITT population will consist of symptomatic patients with biallelic deletion mutations of *SMN1* (exon 7/8 common homozygous deletions) and 2 copies of *SMN2* without the known gene modifier mutation (c.859G>C) who receive an IV infusion of AVXS-101 at less than 180 days of age. All primary and secondary efficacy analyses will be conducted on the ITT population.

#### 14.1.1.2.2. Ability to Thrive ITT Population

The ability to thrive ITT population will consist of symptomatic patients with biallelic deletion mutations of *SMN1*, 2 copies of *SMN2* without the genetic modifier (c.859G>C), intact swallowing and receiving no enteral (mechanical) nutrition at baseline, who receive an IV

Investigational Product: AVXS-101


infusion of AVXS-101 and have at least one post-baseline efficacy evaluation. This population will be utilized to calculate the proportion of patients with the ability to thrive.

#### 14.1.1.3. Efficacy Completers Population

The efficacy completers analysis population will consist of:

- All treated patients who reach 14 months of age, OR
- All treated patients who meet discontinuation criteria, discontinue the trial due to an AE or death

## 14.1.1.4. All Enrolled Population

The all enrolled population will consist all patients who receive an IV infusion of AVXS-101. Analyses of endpoints in this population are considered descriptive.

### 14.1.1.5. Safety Population

The safety analysis population will consist of all patients who receive an IV infusion of AVXS-101. All safety analyses will be conducted on the safety analysis population.

# **14.2.** Sample Size Calculation

The current trial will enroll 30 patients. (Babies who are in screening and meet eligibility criteria for the study at the time the enrollment target is met may be enrolled upon approval of the sponsor.) At least 25 symptomatic patients, ITT population, will have biallelic deletion mutations of *SMN1*, 2 copies of *SMN2* and without the genetic modifier (c.859G>C), ensuring a reasonably robust safety database at the time of the Marketing Authorization Application submission. The trial power is based upon efficacy analysis of the ITT population.

Based upon widely cited natural history of the disease (PNCR) [21], it is expected that no patients in this population would be expected to attain the ability to sit without support or accomplish other developmental milestones (rolling over, standing, walking) prior to reaching 18 months of age. Assuming that the true response rate for the primary endpoint is actually zero (or as low as 0.1%) in the population of interest of the historical control, the primary efficacy endpoint hypothesis is:

**Ho**:  $p_{AVXS-101} = 0.1\%$  versus the alternative

**Ha**: pAVXS-101 > 0.1%,

where *pp* is the proportion of sitting without support for at least 10 seconds up to and including the 18-month trial visit.

Based upon preliminary results from the completed Phase 1 clinical trial AVXS-101-CL-101, at least 50% of treated symptomatic patients with 2 copies of *SMN2* and without the genetic modifier (c.859G>C) are expected to achieve the primary efficacy endpoint of sitting without support for at least 10 seconds up to and including the 18-month trial visit. With the assumption for the true response rate of AVXS-101 being in the range of 20% - 50%, a sample size of 25

Investigational Product: AVXS-101


patients would provide power of greater than 95% to detect a significant difference with  $\alpha = 0.025$  using a 1-sided exact test for a binomial proportion.

Investigational Product: AVXS-101


The secondary efficacy endpoint hypothesis:

**Ho**: pAVXS-101 = pPNCR

versus the alternative

**Ha**:  $pAVXS-101 \neq pPNCR$ 

where pp is the proportion patients of surviving at 14 months of age.

Based upon preliminary results from the same completed Phase 1 clinical trial AVXS-101, at least 80% of treated symptomatic patients with 2 copies of *SMN2* and without the genetic modifier (c.859G>C) are expected to achieve secondary efficacy endpoint of survival at or beyond 14 months of age (based upon the definition of survival outlined above). It is anticipated that 75% of patients in the PNCR population would not survive beyond 13.6 months of age, and that these control patients will represent a 25% survival rate based upon the natural history of the disease. Given this efficacy, a sample size of 25 patients would provide power of >90% to detect a significant difference with  $\alpha = 0.05$  using a 2-sided Fisher's Exact test, as comparing to those control patients with age and gender-matched selected from existing natural history data sets [21], [45].

# 14.3. Efficacy Analysis

#### 14.3.1. General Considerations

This trial will compare the activity of AVXS-101 administered IV versus the natural observational results from PNCR [24] in terms of sitting without support and survival rate.

The analysis of the primary and secondary efficacy endpoints will be performed for the ITT population, and efficacy completers populations. The analysis based on the ITT population will be considered as the primary analysis.

Unless otherwise specified, the baseline measurement is defined as the last non-missing measurement collected prior to or on the day of gene replacement therapy infusion (i.e., on or before Day 1 visit).

#### 14.3.2. Primary and Secondary Efficacy Analysis

Primary and secondary efficacy analyses will be based on ITT population, those symptomatic patients with biallelic Exon 7/8 deletion mutations of *SMN1*, and 2 copies of *SMN2* without the genetic modifier (c.859G>C). These analyses are to test the superiority of AVXS-101 to the results from natural observation trial [24].

The primary efficacy hypothesis to be tested is:

**Ho**: pAvxs-101 = 0.1%

versus the alternative

**Ha**: pAVXS-101 > 0.1%,

where pp is the proportion of sitting without support for at least 10 seconds up to and including the 18 months of age visit, of the ITT population.

The secondary efficacy hypothesis to be tested is:

**Ho**:  $p_{AVXS-101} = p_{PNCR}$ 

versus the alternative

**Ha**: pAVXS-101  $\neq pP$ NCR

where pp is the proportion surviving at 14 months of age in ITT population.

One-sided exact binomial tests (alpha level of 0.025) will be executed for the primary efficacy analysis in the ITT population. For the secondary endpoint, a 2-sided Fisher's Exact test will be used to compare the ITT population with patients from the PNCR natural history trial data-set.

A sensitivity analysis will be conducted by repeating the primary efficacy analysis on the efficacy completers analysis population.

# 14.4. Safety Analysis

Safety will be assessed through the incidence and severity of AEs, vital sign assessments, cardiac assessments, laboratory evaluations (chemistry, hematology, immunology, urinalysis), physical examinations, and use of concomitant medications. Adverse events will be coded in accordance with the most current version of the MedDRA coding dictionary.

Safety analyses will be conducted on safety population.

## 14.4.1. Hy's Law Criteria

In order to assess hepatotoxicity, all elevations in liver transaminases are evaluated using Hy's Law criteria as these help to determine the risk of drug induced liver injury. All elevations in liver transaminases will be assessed against these criteria. Hy's Law cases have the following key components:

- 1. Subjects showing ALT or AST elevations, greater than 3xULN, combined with serum TBL to ≥2xULN, without initial findings of cholestasis (elevated serum ALP);
- 2. No other reason can be found to explain the combination of increased ALT or AST and TBL, such as viral hepatitis A, B, or C, pre-existing or acute liver disease, or another drug capable of causing the observed injury [48].


# 15. DATA SAFETY MONITORING BOARD/DATA MONITORING COMMITTEE

The DSMB/DMC is an independent multidisciplinary group consisting of clinicians and a biostatistician that, collectively, have experience in the management of patients with SMA Type 1 and other diseases, and in the conduct and monitoring of randomized clinical studies with interim analyses. The DSMB/DMC will be chartered to oversee the safety of patients during the conduct of the trial and will act in an advisory capacity to AveXis. A detailed description of the DSMB/DMC, its role in this trial, and the timing of the scheduled reviews will be described in a DSMB/DMC Charter.

The DSMB/DMC will routinely convene on a quarterly basis to review emerging safety data from the trial. Following each meeting, the DSMB/DMC will make a recommendation as to whether or not the accumulated safety data warrants a suspension or discontinuation of the trial, a modification to the trial, or any additional comments or recommendations related to safety. The DSMB/DMC will prepare and provide minutes of their meetings to AveXis who will provide copies to the regulatory authorities as appropriate.


## 16. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 16.1. Trial Monitoring

Before an investigational site can enter a patient into the trial, a representative of AveXis will visit the investigational trial site to:

- Determine the adequacy of the facilities
- Discuss with the Investigator(s) and other personnel their responsibilities with regard to protocol adherence, and the responsibilities of AveXis or its representatives. This will be documented in a Clinical Trial Agreement between AveXis and the Investigator.

During the trial, a monitor from AveXis or representative will have regular contacts with the investigational site, for the following:

- Provide information and support to the Investigator(s)
- Confirm that facilities remain acceptable
- Confirm that the investigational team is adhering to the protocol, that data are being accurately recorded in the case report forms, and that investigational product accountability checks are being performed
- Perform source data verification. This includes a comparison of the data in the case report forms with the patient's medical records at the hospital or practice, and other records relevant to the trial. This will require direct access to all original records for each patient (e.g., clinic charts, electronic medical records)
- Record and report any protocol deviations not previously sent to AveXis
- Confirm AEs and SAEs have been properly documented on eCRFs and confirm any SAEs have been forwarded to AveXis and those SAEs that met criteria for reporting have been forwarded to the IRB/IEC.

The monitor will be available between visits if the Investigator(s) or other staff needs information or advice.

In the event of unforeseen catastrophe or other, serious situation (such as the COVID-19 pandemic) that occurs during the study, which limits or prevents on-site visits, remote site monitoring visits may be conducted. This should not include remote source data verification (SDV), unless in exceptional circumstances, depending upon local regulations and prior informed consent having been obtained from participating subjects.

# 16.2. Audits and Inspections

Authorized representatives of AveXis, a regulatory authority, an IRB/IEC may visit the site to perform audits or inspections, including source data verification. The purpose of an AveXis audit or inspection is to systematically and independently examine all trial-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, Good Clinical Practice (GCP)

Investigational Product: AVXS-101


guidelines of the International Council for Harmonization (ICH), and any applicable regulatory requirements. The Investigator should contact AveXis immediately if contacted by a regulatory agency about an inspection.

# 16.3. Institutional Biosafety Committee

As this trial involves gene therapy, the Principal Investigator must obtain approval/favorable opinion for the investigation from a designated institutional or independent biosafety committee in accordance with institutional requirements and/or guidelines.

# 16.4. Institutional Review Board/Independent Ethics Committee

The Principal Investigator must obtain IRB/IEC approval for the investigation (see Section 18.1). Initial IRB/IEC approval, and all materials approved by the IRB/IEC for this trial including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.


# 17. QUALITY CONTROL AND QUALITY ASSURANCE

Qualified individuals designated by the Sponsor will monitor all aspects of the study according to GCP, standard operating procedures (SOPs), and for compliance with applicable government regulations. Please see Section 16.1 for more details regarding the quality control and monitoring process. AveXis may also conduct a quality assurance audit any time during or after the completion of the study. Please see Section 16.2 for more details regarding the audit process.

The Investigator agrees to allow these Sponsor representatives direct access to the clinical data and supplies, dispensing and storage areas and if requested, agrees to cooperate fully or assist the Sponsor representative. The Investigator and staff are responsible for being present or available for consultation during routinely scheduled site visits conducted by the Sponsor or its designees.

Noncompliance with the protocol, ICH, GCP, or local regulatory requirements by an Investigator, site staff, or representatives of the Sponsor will lead to prompt action by the Sponsor to secure compliance. Continued noncompliance may result in termination of the corresponding party's involvement in the study. The IRB/IEC and relevant regulatory authority will also be informed.

To ensure compliance with Good Clinical Practices and all applicable regulatory requirements, AveXis may conduct a quality assurance audit. Please see Section 16.2 for more details regarding the audit process.


## 18. ETHICS

#### 18.1. Ethics Review

The final trial protocol, including the final version of the Informed Consent Form, must be approved or given a favorable opinion in writing by an IRB/IEC, as appropriate. The Investigator must submit written approval to AveXis before he or she can enroll any patient into the trial.

The Principal Investigator is responsible for informing the IRB/IEC of any amendment to the protocol in accordance with local requirements. In addition, the IRB/IEC must approve all advertising used to recruit patients for the trial. The protocol must be re-approved by the IRB/IEC upon receipt of amendments and annually, as local regulations require.

The Principal Investigator is also responsible for providing the IRB with reports of any reportable serious adverse drug reactions from any other trial conducted with the investigational product. AveXis or designee will provide this information to the Principal Investigator.

Progress reports and notifications of serious adverse drug reactions will be provided to the IRB or IEC according to local regulations and guidelines.

Initial IRB/IEC approval, and all materials approved by the IRB/IEC for this trial including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

#### 18.2. Ethical Conduct of the Trial

The trial will be performed in accordance with ethical principles that have their origin in the Declaration of Helsinki (Appendix 7) and are consistent with ICH/GCP, applicable regulatory requirements.

#### 18.3. Written Informed Consent

The Principal Investigator(s) at each center will ensure that the parent(s)/legal guardian(s) are given full and adequate oral and written information about the nature, purpose, possible risk and benefit of the trial. The parent(s)/legal guardian(s) must also be notified that they are free to discontinue the patient from the trial at any time. The parent(s)/legal guardian(s) should be given the opportunity to ask questions and allowed time to consider the information provided.

The signed and dated informed consent must be obtained before conducting any trial procedures.

The Principal Investigator(s) must maintain the original, signed Informed Consent Form. A copy of the signed Informed Consent Form must be given to the parent(s)/legal guardian(s).

There will be 3 informed consent forms:

- Parent(s)/legal guardian(s) informed consent form
- Biological mother baseline AAV9 antibody screening informed consent form
- Autopsy informed consent form (see Appendix 2; if the parent(s)/legal guardian(s) decline an autopsy, it will not prevent the patient from participating in the trial)

Investigational Product: AVXS-101


In the event of unforeseen catastrophe or other, serious situation (such as the COVID-19 pandemic) that occurs during the study, the ability to obtain a standard written informed consent may be challenged due to limits that prevent an on-site visit. In this situation, the Investigator may conduct the informed consent discussion remotely (e.g. telephone, videoconference). Guidance issued by local regulatory bodies on this aspect prevail and must be implemented and appropriately documented (e.g. the presence of an impartial witness, sign/dating separate ICFs by trial participant and person obtaining informed consent; a video or other recording of the consent process and affirmation of consent may be considered to supplement the documentation of obtaining consent, if allowable by local regulations etc.).


#### 19. DATA HANDLING AND RECORDKEEPING

## 19.1. Electronic Case Report Forms

Adequate and accurate case records will be maintained, and all relevant observations and data related to the trial will be recorded. This will include medical history/ physical examination, hematology, clinical chemistry and serology results, a check list of inclusion and exclusion criteria, product administration, and a record of sample collection, hemodynamic measurements, clinical assessments, AEs, and final evaluation.

Electronic CRFs will be used in this trial. The eCRF will be electronically signed and dated by the Principal Investigator or his designee after his/her review. After the completion of the trial, completed eCRFs will be retained in the archives.

Completed eCRFs will be reviewed by the trial monitor against the source documentation for accuracy and completeness. Once signed by the Investigator, the monitor will transmit the completed eCRFs to data management for data validation and database analysis.

# 19.2. Inspection of Records

AveXis or designee will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the trial. The Investigator agrees to allow the monitor to inspect the product storage area, trial product stocks, product accountability records, patient charts and trial source documents, and other records relative to trial conduct.

## 19.3. Retention of Records

All primary data that are a result of the original observations and activities of the trial and that are necessary for the reconstruction and evaluation of any trial report will be retained in a secure archive at the trial site for a period not < 2 years after the last approval of a marketing application in an ICH region, and until there are no pending or contemplated marketing applications in an ICH region, or until at least 2 years have lapsed since the formal discontinuation of the clinical development of the investigational product. All country/region specific requirements that may be more stringent than the 2 years included in ICH shall be followed.

The site will maintain essential documents as required by ICH-GCP. The site must keep these documents available for review by the Sponsor, IRB/IEC, and/or regulatory bodies.


## 20. PUBLICATION POLICY

The Investigator is obliged to provide the Sponsor with complete test results and all data derived by the Investigator from the trial. During the trial, only the Sponsor may make trial information available to other trial Investigators or to regulatory agencies, except as required by law or regulation. Except as otherwise allowable in the clinical trial site agreement, any public disclosure (including publicly accessible websites) related to the protocol or trial results, other than trial recruitment materials and/or advertisements, is the sole responsibility of the Sponsor.

The Sponsor may publish any data and information from the trial (including data and information generated by the Investigator) without the consent of the Investigator. Manuscript authorship for any peer-reviewed publication will appropriately reflect contributions to the production and review of the document. All publications and presentations must be prepared in accordance with this section and the Clinical Trial Site Agreement. In the event of any discrepancy between the protocol and the Clinical Trial Site Agreement, the Clinical Trial Site Agreement will prevail.

If the trial is being conducted as part of a multicenter clinical trial, data from all sites participating in the trial will be pooled and analyzed by the Sponsor or the Sponsor's designee. The first publication of the trial results shall be made in conjunction with the results from other trial sites as a multicenter publication. If a multicenter publication is not forthcoming within 24 months of completion of the trial at all sites, the Investigator may publish or present the results generated at his or her site.

The Investigator will provide the Sponsor with a copy of any proposed publication or presentation for review and comment at least 60 days prior to such presentation or submission for publication. The Sponsor shall inform the Investigator in writing of any changes or deletions in such presentation or publication required to protect the Sponsor's confidential and proprietary technical information and to address inaccurate data or inappropriate interpretations in the context of any pooled multicenter results. At the expiration of such 60-day period, the Investigator may proceed with the presentation or submission for publication unless the Sponsor has notified the institution or the Investigator in writing that such proposed publication or presentation discloses the Sponsor's confidential and proprietary technical information. Further, upon the request of the Sponsor, the Investigator will delay the publication or presentation for an additional 90 days to permit the Sponsor to take necessary actions to protect its intellectual property interests.

Investigational Product: AVXS-101


## 21. LIST OF REFERENCES

- 1. Sugarman EA, Nagan N, Zhu H, et al. Pan-ethnic carrier screening and prenatal diagnosis for spinal muscular atrophy: clinical laboratory analysis of >72,400 specimens. *Eur J Hum Genet*. 2012;20(1):27-32.
- 2. Swoboda KJ, Prior TW, Scott CB, et al. Natural history of denervation in SMA: relation to age, *SMN2* copy number, and function. *Ann Neurol.* 2005;57(5):704-712.
- 3. Le TT, McGovern VL, Alwine IE, et al. Temporal requirement for high SMN expression in SMA mice. *Hum Mol Genet*. 2011;20(18):3578-3591.
- 4. Farrar MA, Vucic S, Johnston HM, Kiernan MC. Corticomotoneuronal integrity and adaptation in spinal muscular atrophy. *Arch Neurol*. 2012b;69(4):467-473.
- 5. Riessland M, Ackermann B, Forster A, et al. SAHA ameliorates the SMA phenotype in 2 mouse models for spinal muscular atrophy. *Hum Mol Genet*. 2010;19(8):1492-1506.
- Dayangac-Erden D, Bora-Tatar G, Dalkara S, Demir AS, Erdem-Yurter H. Carboxylic acid derivatives of histone deacetylase inhibitors induce full length SMN2 transcripts: a promising target for spinal muscular atrophy therapeutics. Arch Med Sci. 2011;7(2):230-234.
- 7. National Library of Medicine [Available from: www.ClinicalTrials.gov]
- 8. Darbar IA, Plaggert PG, Resende MB, Zanoteli E, Reed UC. Evaluation of muscle strength and motor abilities in children with Type II and III spinal muscle atrophy treated with valproic acid. *BMC Neurol*. 2011;11:36.
- 9. Mercuri E, Bertini E, Iannaccone ST. Childhood spinal muscular atrophy: controversies and challenges. *Lancet Neurol.* 2012;11(5):443-452.
- 10. Kolb SJ, Kissel JT. Spinal muscular atrophy: a timely review. *Arch Neurol.* 2011;68(8):979-984.
- 11. Lefebvre S, Burglen L, Reboullet S, Clermont O, Burlet P, Viollet L, et al. Identification and characterization of a spinal muscular atrophy-determining gene. *Cell*. 1995;80(1):155-164.
- 12. Lorson CL, Hahnen E, Androphy EJ, Wirth B. A single nucleotide in the SMN gene regulates splicing and is responsible for spinal muscular atrophy. *Proc Natl Acad Sci USA*. 1999;96(11):6307-6311.
- 13. Monani UR, Lorson CL, Parsons DW, Prior TW, Androphy EJ, Burghes AH et al. A single nucleotide difference that alters splicing patterns distinguishes the SMA gene *SMN1* from the copy gene *SMN2*. *Hum Mol Genet*. 1999;8(7):1177-1183.
- 14. Lefebvre S, Burlet P, Liu Q, et al. Correlation between severity & SMN protein level in spinal muscular atrophy. *Nat Genet*. 1997;16(3):264-269.
- 15. Park GH, Kariya S, Monani UR. Spinal muscular atrophy: new and emerging insights from model mice. *Curr Neurol Neurosci Rep.* 2010;10(2):108-117.

Investigational Product: AVXS-101

- 16. Feldkotter M, Schwarzer V, Wirth R, Wienker TF, Wirth B. Quantitative analyses of *SMN1* and *SMN2* based on real-time lightCycler PCR: fast and highly reliable carrier testing and prediction of severity of spinal muscular atrophy. *Am J Hum Genet*. 2002;70(2):358-368.
- 17. Prior TW, Krainer AR, Hua Y, et al. A positive modifier of spinal muscular atrophy in the *SMN2* gene. *Am J Hum Genet.* 2009;85:408-413.
- 18. Farrar MA, Vucic S, Johnston HM, et al. Pathophysiological insights derived by natural history and motor function of spinal muscular atrophy. *J Pediatr*. 2013;162(1):155-159.
- 19. Foust KD, Wang X, McGovern VL, et al. Rescue of the spinal muscular atrophy phenotype in a mouse model by early postnatal delivery of SMN. *Nat Biotechnol*. 2010;28(3):271-274.
- 20. Hinderer C, Katz N, Buza EL, et al. Severe toxicity in nonhuman primates and piglets following high-dose intravenous administration of an adeno-associated virus vector expressing human SMN. *Hum Gene Ther.* 2018 Mar;29(3):285-298.
- 21. Hordeaux J, Hinderer C, Goode T, et al. Toxicology study of intra-cisterna magna adenoassociated virus 9 expressing human alpha-L-iduronidase in rhesus macaques. *Mol Ther Methods Clin Dev.* 2018 Jul 14;10:79-88.
- 22. Butchbach ME, Edwards JD, Burghes AH. Abnormal motor phenotype in the SMNDelta7 mouse model of spinal muscular atrophy. *Neurobiol Dis.* 2007;27(2):207-219.
- 23. Finkel RS, McDermott MP, Kaufmann P, et al. Observational trial of spinal muscular atrophy Type I and implications for clinical trials. *Neurol*. 2014;83(9):810-817.
- 24. Swoboda KJ, Prior TW, Scott CB, et al. Natural history of denervation in SMA: relation to age, SMN2 copy number, and function. *Ann Neurol*. 2005;57(5):704-12.
- 25. AVXS-101 Investigator's Brochure version 6.0. 17 September 2019. AveXis, Inc., Bannockburn, IL.
- 26. Narver HL, Kong L, Burnett BG, et al. Sustained improvement of spinal muscular atrophy mice treated with trichostatin A plus nutrition. *Ann Neurol.* 2008;64(4)465-470.
- 27. Paes BA, Mitchell I, Banerji A, Lanctot KL, Langley JM. A decade of respiratory syncytial virus epidemiology and prophylaxis: translating evidence into everyday practice. *Can Respir J.* 2001;18(2): e10-9.
- 28. Nair H, Nokes DJ, Gessner BD, et al. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. *Lancet*, 2010; 375:1545–55.
- 29. Hall CB. Respiratory syncytial virus and parainfluenza virus. *New Engl J Med*. 2001;344:1917-1928.

Investigational Product: AVXS-101

- 30. Palivizumab SmPC. www.ema.europa.eu/en/documents/product-information/synagis-epar-product-information en.pdf. April 6, 2019.
- 31. Finkel RS, Mercuri E, Meyer OH, et al. SMA Care group. Diagnosis and management of spinal muscular atrophy: Part 2: Pulmonary and acute care; medications, supplements and immunizations; other organ systems; and ethics. *Neuromuscul Disord*. 2018;28(3):197-207.
- 32. McCarty DM, Young Jr SM, Samulski RJ. Integration of adeno-associated virus (AAV) and recombinant AAV vectors. *Ann Rev Genet*. 2004;38:819-845.
- 33. Kotin RM, Siniscalco M, Samulski RJ, et al. Site-specific integration by adeno-associated virus. *Proc Natl Acad Sci USA*. 1990;87(6):2211-2215.
- 34. Surosky RT, Urabe M, Godwin SG, et al. Adeno-associated virus Rep proteins target DNA sequences to a unique locus in the human genome. *J Virol*. 1997;71(10):7951-7959.
- 35. Srivastava A and Carter BJ. AAV infection: protection from cancer. *Hum Gene Ther*. 2017;28(4):323-327.
- 36. Favre D, Provost N, Blouin V, et al. "Immediate and long-term safety of recombinant adeno-associated virus injection into the nonhuman primate muscle." *Mol Ther*. 2001;4.6:559-566.
- 37. Afione SA, Conrad CK, Kearns WG, et al. In vivo model of adeno-associated virus vector persistence and rescue. *J Virol.* 1996;70.5:3235-3241.
- 38. Wijnhoven TMA, De Onis M, Oyango AW, Wang T, Bjoerneboe GA, Bhandari N, Lartey A, Al Rashidi B; WHO Multicentre Growth Reference Trial Group. Assessment of gross motor development in the WHO multicenter growth reference trial. *Food Nutr Bull*. 2004;25(1 Suppl 1):S37S45.
- 39. Albers CA, Grieve AJ. Test Review: Bayley, N. (2006). Bayley Scales of Infant and Toddler Development- Third Edition. San Antonio, TX: Harcourt Assessment. *J Psychoeduc Assess*. 2007;25(2):180-198.
- 40. US Department of Health and Human Services. Common Terminology Criteria for Adverse Events (v4.03). Published May 2009 (Revised June 2010).
- 41. Zoorob RJ, Cender D. A different look at corticosteroids. *Am Fam Physician*. 1998;58(2):443-450.
- 42. Onis M. WHO Child Growth Standards based on length/height, weight and age. *Acta Paediatr.* 2006;95.S450:76-85.
- 43. Kroger A, Duchin J, Vazquez M. General Best Practice Guidelines for Immunization (ACIP). www.cdc.gov/vaccines/hcp/acip-recs/general-recs/downloads/general-recs.pdf. Accessed on 2018.
- 44. Palivizumab Summary of Product Characteristics. [https://www.ema.europa.eu/en/documents/product-information/synagis-epar-product-information en.pdf] 2018

Investigational Product: AVXS-101

- 45. Glanzman AM, McDermott MP, Montes J, et al. Validation of the Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND). *Pediatr Phys Ther*. 2011;23(4):322-326.
- 46. Glanzman AM, Mazzone E, Main M, et al. The Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND): test development and reliability. *Neuromusc Disord*. 2010;20(3):155-161.
- 47. Kolb S. Longitudinal results from the NeuroNEXT SMA infant biomarker trial. Presented at: 20th Annual International Spinal Muscular Atrophy Research Group Meeting; June 2016; Anaheim, CA.
- 48. FDA (2009) U.S. Department of Health and Human Services, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER). Guidance for Industry. Drug-Induced Liver Injury: Premarketing Clinical Evaluation; <a href="https://www.fda.gov/downloads/guidances/UCM174090.pdf">https://www.fda.gov/downloads/guidances/UCM174090.pdf</a>.


# 22. APPENDICES

## APPENDIX 1. SCHEDULE OF ASSESSMENTS

| Trial Period | Screen-<br>ing | | • | lacemo | | | | | | | Fo | ollow- | up (Outpa | tient) | Notes | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nominal Study Day (Visit Relative To Dose) | −30 to −2 | -1 | 1 | 2 | 3 | 7 | 14 | 21 | 30 | 44 | 60 (or<br>Month<br>2) | 72 | 90 (or<br>Month 3 | Month<br>4,5,7,8,10,11,13 | Month 6,9,12 | (18 months | Depending on the patient's age at dosing,<br>the duration of participation can vary from |
| Visit According To<br>Months of Age | | | | | | | | | | | | | | 14,16,17 | 15 | of age or ET | approximately 12 months (baby dosed at approximately 6 months of age) to approximately 18 months (baby dosed near |
| Window | | (No W | indow | ·) | | | ± | : <b>2 d</b> a | iys | | (Exce | ept +0 | | days<br>at 14 Months of A | Age) | +0-14 days | birth, "0 months of age"). |
| Informed Consent | Х | | | | | | | | | | | | | | | | See Section 18.3. |
| AVXS-101 Infusion | | | х | | | | | | | | | | | | | | See Section 10.6. Day 1 assessments will be performed prior to the start of gene replacement therapy infusion. |
| BSIDv03/WHO<br>Developmental<br>Milestones (with video) | Х | | | | | | | | Х | | х | | х | Х | х | Х | See Sections 11.1, 11.2.1, 11.2.2 and 11.3. |
| BSIDv03 Gross and Fine<br>Motor Subtests (with<br>video) | Х | | | | | | | | Х | | Х | | Х | Х | х | Х | See Sections 11.1, 11.2.1, 11.2.2 and 11.3. |
| CHOP INTEND (with video) | Х | Х | | | | Х | Х | Х | Х | | Х | | Х | Х | х | l X | See Sections 11.2.3 and 11.3. Patients who achieve 3 consecutive CHOP INTEND scores ≥ 58 will not continue CHOP INTEND assessments. |


| Trial Period | Screen-<br>ing | | e Rep | | | | | | | | Fo | ollow- | up (Outpa | atient) | Notes | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nominal Study Day (Visit Relative To Dose) | -30 to −2 | -1 | 1 | 2 | 3 | 7 | 14 | 21 | 30 | 44 | 60 (or<br>Month<br>2) | 72 | 90 (or<br>Month 3 | Month<br>4,5,7,8,10,11,13 | Month 6,9,12 | (18 months | |
| Visit According To<br>Months of Age | | | | | | | | | | | | | | 14,16,17 | 15 | of age or ET) | approximately 12 months (baby dosed at approximately 6 months of age) to approximately 18 months (baby dosed near |
| Window | | (No W | indow | ·) | | | ± | : <b>2</b> da | ys | | (Exce | ept +0 | | days<br>at 14 Months of A | Age) | +0-14 days | birth, "0 months of age"). |
| Demographic/Medical<br>History | Х | | | | | | | | | | | | | | | 2 | See Section 12.1.1. |
| Physical Exam | Х | | Х | Х | Х | Χ | Χ | Х | Χ | | Х | | Х | Х | Х | Х | See Section 12.1.2. |
| Vital Signs/Weight &<br>Length | X | Х | (X) | х | x | x | X | x | X | | Х | | Х | X | х | Х | See Section 12.1.3. (X): Vital signs will be continuously monitored throughout the infusion of gene replacement therapy and recorded every 15 minutes (+/- 5 minutes) post dose for the first 4 hours after the start of infusion, then every hour (+/- 15 minutes) until 24 hours after the start of infusion. Axillary temperature will be recorded pre- and post-infusion. |
| 12-Lead ECG | Х | | | Х | | | | | Χ | | | | (X) | (X) | (X) | Х | See Sections 12.1.4, 12.1.5, and 12.1.6. |
| Echocardiogram | Х | | | | | | | | Χ | | | | (X) | (X) | (X) | Х | (X): Completed every 3 months, starting at Month 3 until 12 months post-dose. |
| 24-hour Holter Monitor | Х | Х | Х | Х | Χ | | | | Χ | | Х | | (X) | (X) | (X) | Х | |
| Pulmonary Examination | Х | Х | | Х | Х | Х | Χ | Χ | Χ | | Х | | Х | Х | Х | Х | See Section 12.1.7. |
| Swallowing Test | Х | | | | | | | | | | | | | | (X) | (X) | See Section 12.1.8. |


| Trial Period | Screen-<br>ing | | e Repl<br>apy (Ir | | | | | | | | Fo | ollow- | up (Outpa | itient) | | Notes | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nominal Study Day (Visit Relative To Dose) | -30 to -2 | -1 | 1 | 2 | 3 | 7 | 14 | 21 | 30 | 44 | 60 (or<br>Month<br>2) | 72 | 90 (or<br>Month 3 | Month<br>4,5,7,8,10,11,13 | Month 6,9,12 | (18 months | illie dulation of participation can vary more |
| Visit According To<br>Months of Age | | | | | | | | | | | | | | 14,16,17 | 15 | of age or ET) | approximately 12 months (baby dosed at approximately 6 months of age) to approximately 18 months (baby dosed near |
| Window | | (No W | indow | ) | | | ± | : <b>2</b> da | ys | | (Exce | ept +0 | | days<br>at 14 Months of A | lge) | +0-14 days | birth, "0 months of age"). |
| | | | | | | | | | | | | | | | | 20 | (X): Completed every 6 months, starting at<br>Month 6 through the End of Trial at<br>18 months of age. |
| Photograph of Infusion<br>Site | | | (X) | Х | х | х | х | х | х | | | | | | | | See Section 12.1.9. (X): Day 1 infusion site photograph will be performed prior to the start of gene replacement therapy infusion. |
| Hematology/Chemistry<br>/Urinalysis | х | (X) | | х | | х | х | х | х | (X)* | х | (X)* | х | х | х | х | See Sections 12.1.10.1, 12.1.10.2 and 12.1.10.3. (X): Laboratory samples collected on Day -1 to be processed locally, prior to dosing. (X)*: Liver function test (AST, ALT, total bilirubin, direct bilirubin, alkaline phosphatase, GGT) only. |
| CK-MB or Troponin I | Х | | | | | Χ | | | Χ | | Х | | | | Х | Х | See Section 12.1.10.2. |
| Virus Serology | Х | | | | | | | | | | | | | | | | See Section 12.1.10.4. |
| Capillary Blood Gas | | Χ | | Х | | | | | | | | | | | | | See Section 12.1.10.5. |
| Immunological Testing:<br>ELISA (anti-AAV9/SMN<br>Ab) | Х | | | | | х | Х | х | х | | | | | | | | See Section 12.1.10.6. |


| Trial Period | Screen-<br>ing | | • | lacemon-pation | | | | | | | | ollow- | up (Outpa | itient) | Notes | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Nominal Study Day (Visit Relative To Dose) | -30 to −2 | -1 | 1 | 2 | 3 | 7 | 14 | 21 | 30 | 44 | 60 (or<br>Month<br>2) | 72 | 90 (or<br>Month 3 | Month<br>4,5,7,8,10,11,13 | Month 6,9,12 | (18 months | Depending on the patient's age at dosing,<br>the duration of participation can vary from |
| Visit According To<br>Months of Age | | | | | | | | | | | | | | 14,16,17 | 15 | of age or ET | approximately 12 months (baby dosed at approximately 6 months of age) to approximately 18 months (baby dosed near |
| Window | | (No W | indow | ·) | | | ± | ± 7 days<br>± 2 days<br>(Except +0–14 days at 14 Months of Age) | | | | +0-14 days | birth, "0 months of age"). | | | | |
| AAV9 Ab Screen in<br>Biological Mother | Х | | | | | | | | | | | | | | | 2 | See Section 12.1.10.7. |
| Blood for Diagnostic<br>Confirmation Testing | Х | | | | | | | | | | | | | | | 40 | See Section 12.1.10.8. |
| Saliva, Urine, and Stool<br>Samples (for viral<br>shedding) | Х | | | (X) | (X) | х | х | х | х | | | | | | | | See Section 12.1.10.9. (X): Collected within 24 and 48 hours post dose. |
| Prophylactic<br>Prednisolone | | х | х | х | х | х | х | х | х | (X) | (X) | | | | | | See Section 9.2.1. (X): After 30 days, prednisolone (or equivalent glucocorticoid) can be tapered for patients whose ALT values, and AST values are below the threshold. |
| Adverse Events | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | See Section 13. |
| Prior and Concomitant<br>Medications | Collected from 2 weeks before gene replacement therapy until End of Trial visit | | | | | | | | | | | | | | | | |

Ab = antibody; ALT = alanine aminotransferase; AST = aspartate aminotransferase; BSIDv03 = Bayley Scales of Infant and Toddler Development version 3;

CBC = complete blood count; CHOP INTEND = Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders; CK-MB = Creatinine kinase-muscle/brain;

ECG = electrocardiogram; ELISA = enzyme-linked immunosorbent assay; ET = early termination; GGT = gamma glutamyl transferase; IRB = Institutional Review Board; LFT = liver function tests; WHO = World Health Organization


#### APPENDIX 2. POST-MORTEM TISSUE AND ORGAN COLLECTION PLAN

Post-mortem tissue/organ collection and autopsy, where possible, will be requested for any patient who receives gene replacement therapy. The autopsy and tissue collection will be performed by the clinical site local pathologist or a contracted vendor who may deploy a pathology assistant to the funeral home, hospital, or other applicable location to perform the tissue and organ collection. Standard autopsy incisions will be used to perform the procedures.

During the procedure, multiple tissues along with the entire spinal cord will be collected for research purposes, including up to 7 sections or pieces from each organ and each region of the spinal cord. Upon collection, these tissue samples will be provided to AveXis for analysis.

Tissue analysis will be done to determine whether the vector transduced the expected motor neurons and if the SMN gene was expressed. These results will demonstrate whether the vector delivered the therapeutic gene as expected. Tissue samples collected will also be available for histology and immunohistochemistry, allowing the state of the motor neurons and muscles to be examined.

Specifically, tissue samples from the spinal cord, muscles, and organs will be collected as indicated in Table 5. Tissue samples will be frozen or fixed (e.g., 2% paraformaldehyde) for appropriate analysis.

Families may be asked to consent to authorize tissue collection prior to any sign of moribund or death by the clinical team conducting the trial. Declining the post-mortem tissue and organ collection will not prevent patients from participating in the trial.

**Table 5: Tissue Sample for Analysis** 

| Brain | Spinal Cord | Muscles | Organs |
|---|---|---|---|
| Motor cortex | Cervical spinal cord | Diaphragm | Spleen |
| Layer 5 motor cortex | Thoracic spinal cord | #6/#7 Rib with intercostal muscle and nerve | Kidney |
| Brain stem | Lumbar spinal cord | Psoas muscle | Small intestine |
| | Sacral spinal cord | | Large intestine |
| | Dorsal root | | Pancreas |
| | Cervical level | | Stomach |
| | Ventral root | | Lung |
| | Cervical level | | Heart |
| | DRG root | | Liver |

Investigational Product: AVXS-101

| Cervical level | Inguinal lymph node |
|---------------------|---------------------|
| Cerebrospinal fluid | Gonads |



Investigational Product: AVXS-101



Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101



Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101



Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101

Protocol Version 7.0/Amendment 6/25 Jun 2020 Investigational Product: AVXS-101

AVXS-101-CL-302 AveXis, Inc.

Investigational Product: AVXS-101
Investigational Product: AVXS-101

AVXS-101-CL-302 AveXis, Inc.

Investigational Product: AVXS-101

Investigational Product: AVXS-101



Investigational Product: AVXS-101



Investigational Product: AVXS-101

Investigational Product: AVXS-101

Investigational Product: AVXS-101


# APPENDIX 4. PERFORMANCE CRITERIA FOR BAYLEY SCALES INFANT AND TODDLER DEVELOPMENT (VERSION 3) DEVELOPMENTAL MILESTONES

| Developmental Milestone |
|------------------------------------------------------------|
| Head Control – Gross Motor Subtest<br>Item #4 |
| Rolls from Back to Sides – Gross<br>Motor Subtest Item #20 |
| Sits Without Support – Gross Motor<br>Subtest Item #26 |
| Stands With Assistance – Gross Motor<br>Subtest Item #33 |
| Crawls – Gross Motor Subtest Item<br>#34 |
| Pulls to Stand – Gross Motor Subtest<br>Item #35 |
| Walks With Assistance – Gross Motor<br>Subtest Item #37 |
| Stands Alone – Gross Motor Subtest<br>Item #40 |
| Walks Alone – Gross Motor Subtest<br>Item #42 |

AVXS-101-CL-302 AveXis, Inc.


#### **APPENDIX 5.** PERFORMANCE CRITERIA FOR WORLD HEALTH **ORGANIZATION (WHO) DEVELOPMENTAL MILESTONES**



Source: World Health Organization Multicentre Growth Reference Trial Group [38]

Investigational Product: AVXS-101


# APPENDIX 6. CHOP INTEND



Investigational Product: AVXS-101

Investigational Product: AVXS-101




# APPENDIX 7. DECLARATION OF HELSINKI: ETHICAL PRINCIPLES FOR MEDICAL RESEARCH INVOLVING HUMAN SUBJECTS

Adopted by the 18<sup>th</sup> WMA General Assembly, Helsinki, Finland, June 1964 and amended by the: 29<sup>th</sup> WMA General Assembly, Tokyo, Japan, October 1975

35<sup>th</sup> WMA General Assembly, Venice, Italy, October 1983

41st WMA General Assembly, Hong Kong, September 1989

48<sup>th</sup> WMA General Assembly, Somerset West, Republic of South Africa, October 1996

52<sup>nd</sup> WMA General Assembly, Edinburgh, Scotland, October 2000

53rd WMA General Assembly, Washington DC, USA, October 2002 (Note of Clarification added)

55<sup>th</sup> WMA General Assembly, Tokyo, Japan, October 2004 (Note of Clarification added)

59th WMA General Assembly, Seoul, Republic of Korea, October 2008

64<sup>th</sup> WMA General Assembly, Fortaleza, Brazil, October 2013

1. The World Medical Association (WMA) has developed the Declaration of Helsinki as a statement of ethical principles for medical research involving Human subjects, including research on identifiable human material and data.

The Declaration is intended to be read as a whole and each of its constituent paragraphs should be applied with consideration of all other relevant paragraphs.

2. Consistent with the mandate of the WMA, the Declaration is addressed primarily to physicians. The WMA encourages others who are involved in medical research involving Human subjects to adopt these principles.

#### **General Principles**

- 3. The Declaration of Geneva of the WMA binds the physician with the words, "The health of my patient will be my first consideration," and the International Code of Medical Ethics declares that, "A physician shall act in the patient's best interest when providing medical care."
- 4. It is the duty of the physician to promote and safeguard the health, well-being and rights of patients, including those who are involved in medical research. The physician's knowledge and conscience are dedicated to the fulfilment of this duty.
- 5. Medical progress is based on research that ultimately must include studies involving Human subjects.

Investigational Product: AVXS-101


- 6. The primary purpose of medical research involving Human subjects is to understand the causes, development and effects of diseases and improve preventive, diagnostic and therapeutic interventions (methods, procedures and treatments). Even the best proven interventions must be evaluated continually through research for their safety, effectiveness, efficiency, accessibility and quality.
- 7. Medical research is subject to ethical standards that promote and ensure respect for all Human subjects and protect their health and rights.
- 8. While the primary purpose of medical research is to generate new knowledge, this goal can never take precedence over the rights and interests of individual research patients.
- 9. It is the duty of physicians who are involved in medical research to protect the life, health, dignity, integrity, right to self-determination, privacy, and confidentiality of personal information of research patients. The responsibility for the protection of research patients must always rest with the physician or other health care professionals and never with the research patients, even though they have given consent.
- 10. Physicians must consider the ethical, legal and regulatory norms and standards for research involving Human subjects in their own countries as well as applicable international norms and standards. No national or international ethical, legal or regulatory requirement should reduce or eliminate any of the protections for research patients set forth in this Declaration.
- 11. Medical research should be conducted in a manner that minimizes possible harm to the environment.
- 12. Medical research involving Human subjects must be conducted only by individuals with the appropriate ethics and scientific education, training and qualifications. Research on patients or healthy volunteers requires the supervision of a competent and appropriately qualified physician or other health care professional.
- 13. Groups that are underrepresented in medical research should be provided appropriate access to participation in research.
- 14. Physicians who combine medical research with medical care should involve their patients in research only to the extent that this is justified by its potential preventive, diagnostic or therapeutic value and if the physician has good reason to believe that participation in the research trial will not adversely affect the health of the patients who serve as research patients.
- 15. Appropriate compensation and treatment for patients who are harmed as a result of participating in research must be ensured.

#### **Risks, Burdens and Benefits**

Investigational Product: AVXS-101


- 16. In medical practice and in medical research, most interventions involve risks and burdens. Medical research involving Human subjects may only be conducted if the importance of the objective outweighs the risks and burdens to the research patients.
- 17. All medical research involving Human subjects must be preceded by careful assessment of predictable risks and burdens to the individuals and groups involved in the research in comparison with foreseeable benefits to them and to other individuals or groups affected by the condition under investigation.
  - Measures to minimize the risks must be implemented. The risks must be continuously monitored, assessed and documented by the researcher.
- 18. Physicians may not be involved in a research trial involving Human subjects unless they are confident that the risks have been adequately assessed and can be satisfactorily managed.

When the risks are found to outweigh the potential benefits or when there is conclusive proof of definitive outcomes, physicians must assess whether to continue, modify or immediately stop the trial.

#### **Vulnerable Groups and Individuals**

19. Some groups and individuals are particularly vulnerable and may have an increased likelihood of being wronged or of incurring additional harm.

All vulnerable groups and individuals should receive specifically considered protection.

20. Medical research with a vulnerable group is only justified if the research is responsive to the health needs or priorities of this group and the research cannot be carried out in a non-vulnerable group. In addition, this group should stand to benefit from the knowledge, practices or interventions that result from the research.

#### **Scientific Requirements and Research Protocols**

- 21. Medical research involving Human subjects must conform to generally accepted scientific principles, be based on a thorough knowledge of the scientific literature, other relevant sources of information, and adequate laboratory and, as appropriate, animal experimentation. The welfare of animals used for research must be respected.
- 22. The design and performance of each research trial involving Human subjects must be clearly described and justified in a research protocol.

The protocol should contain a statement of the ethical considerations involved and should indicate how the principles in this Declaration have been addressed. The protocol should include information regarding funding, Sponsors, institutional affiliations, potential conflicts of interest, incentives for patients and information regarding provisions for treating and/or compensating patients who are harmed as a consequence of participation in the research trial.

Investigational Product: AVXS-101


In clinical trials, the protocol must also describe appropriate arrangements for post-trial provisions.

#### **Research Ethics Committees**

23. The research protocol must be submitted for consideration, comment, guidance and approval to the concerned research ethics committee before the trial begins. This committee must be transparent in its functioning, must be independent of the researcher, the Sponsor and any other undue influence and must be duly qualified. It must take into consideration the laws and regulations of the country or countries in which the research is to be performed as well as applicable international norms and standards but these must not be allowed to reduce or eliminate any of the protections for research patients set forth in this Declaration.

The committee must have the right to monitor ongoing studies. The researcher must provide monitoring information to the committee, especially information about any serious adverse events. No amendment to the protocol may be made without consideration and approval by the committee. After the end of the trial, the researchers must submit a final report to the committee containing a summary of the trial's findings and conclusions.

#### **Privacy and Confidentiality**

24. Every precaution must be taken to protect the privacy of research patients and the confidentiality of their personal information.

#### **Informed Consent**

- 25. Participation by individuals capable of giving informed consent as patients in medical research must be voluntary. Although it may be appropriate to consult family members or community leaders, no individual capable of giving informed consent may be enrolled in a research trial unless he or she freely agrees.
- 26. In medical research involving Human subjects capable of giving informed consent, each potential subject must be adequately informed of the aims, methods, sources of funding, any possible conflicts of interest, institutional affiliations of the researcher, the anticipated benefits and potential risks of the trial and the discomfort it may entail, post-trial provisions and any other relevant aspects of the trial. The potential subject must be informed of the right to refuse to participate in the trial or to withdraw consent to participate at any time without reprisal. Special attention should be given to the specific information needs of individual potential patients as well as to the methods used to deliver the information.

After ensuring that the potential subject has understood the information, the physician or another appropriately qualified individual must then seek the potential subject's freely-given informed consent, preferably in writing. If the consent cannot be expressed in writing, the non-written consent must be formally documented and witnessed.

Investigational Product: AVXS-101


All medical research patients should be given the option of being informed about the general outcome and results of the trial.

- 27. When seeking informed consent for participation in a research trial the physician must be particularly cautious if the potential subject is in a dependent relationship with the physician or may consent under duress. In such situations the informed consent must be sought by an appropriately qualified individual who is completely independent of this relationship.
- 28. For a potential research subject who is incapable of giving informed consent, the physician must seek informed consent from the legally authorized representative. These individuals must not be included in a research trial that has no likelihood of benefit for them unless it is intended to promote the health of the group represented by the potential subject, the research cannot instead be performed with persons capable of providing informed consent, and the research entails only minimal risk and minimal burden.
- 29. When a potential research subject who is deemed incapable of giving informed consent is able to give assent to decisions about participation in research, the physician must seek that assent in addition to the consent of the legally authorized representative. The potential subject's dissent should be respected.
- 30. Research involving patients who are physically or mentally incapable of giving consent, for example, unconscious patients, may be done only if the physical or mental condition that prevents giving informed consent is a necessary characteristic of the research group. In such circumstances the physician must seek informed consent from the legally authorized representative. If no such representative is available and if the research cannot be delayed, the trial may proceed without informed consent provided that the specific reasons for involving patients with a condition that renders them unable to give informed consent have been stated in the research protocol and the trial has been approved by a research ethics committee. Consent to remain in the research must be obtained as soon as possible from the subject or a legally authorized representative.
- 31. The physician must fully inform the patient which aspects of their care are related to the research. The refusal of a patient to participate in a trial or the patient's decision to withdraw from the trial must never adversely affect the patient-physician relationship.
- 32. For medical research using identifiable human material or data, such as research on material or data contained in biobanks or similar repositories, physicians must seek informed consent for its collection, storage and/or reuse. There may be exceptional situations where consent would be impossible or impracticable to obtain for such research. In such situations the research may be done only after consideration and approval of a research ethics committee.

#### Use of Placebo

33. The benefits, risks, burdens and effectiveness of a new intervention must be tested against those of the best proven intervention(s), except in the following circumstances:

Investigational Product: AVXS-101


Where no proven intervention exists, the use of placebo, or no intervention, is acceptable; or where for compelling and scientifically sound methodological reasons the use of any intervention less effective than the best proven one, the use of placebo, or no intervention is necessary to determine the efficacy or safety of an intervention and the patients who receive any intervention less effective than the best proven one, placebo, or no intervention will not be subject to additional risks of serious or irreversible harm as a result of not receiving the best proven intervention. Extreme care must be taken to avoid abuse of this option.

#### **Post-Trial Provisions**

34. In advance of a clinical trial, Sponsors, researchers and host country governments should make provisions for post-trial access for all patients who still need an intervention identified as beneficial in the trial. This information must also be disclosed to patients during the informed consent process.

#### **Research Registration and Publication and Dissemination of Results**

- 35. Every research trial involving Human subjects must be registered in a publicly accessible database before recruitment of the first subject.
- 36. Researchers, authors, Sponsors, editors and publishers all have ethical obligations with regard to the publication and dissemination of the results of research. Researchers have a duty to make publicly available the results of their research on Human subjects and are accountable for the completeness and accuracy of their reports. All parties should adhere to accepted guidelines for ethical reporting. Negative and inconclusive as well as positive results must be published or otherwise made publicly available. Sources of funding, institutional affiliations and conflicts of interest must be declared in the publication. Reports of research not in accordance with the principles of this Declaration should not be accepted for publication.

#### **Unproven Interventions in Clinical Practice**

37. In the treatment of an individual patient, where proven interventions do not exist or other known interventions have been ineffective, the physician, after seeking expert advice, with informed consent from the patient or a legally authorized representative, may use an unproven intervention if in the physician's judgement it offers hope of saving life, reestablishing health or alleviating suffering. This intervention should subsequently be made the object of research, designed to evaluate its safety and efficacy. In all cases, new information must be recorded and, where appropriate, made publicly available.


# **APPENDIX 8. SUMMARY OF CHANGES**

The section below describes the changes incorporated into this version of the protocol.




### **AVXS-101**

# AVXS-101-CL-302

**Protocol Title:** Phase 3, Open-Label, Single-Arm, Single-Dose Gene

Replacement Therapy Clinical Trial for Patients with Spinal Muscular Atrophy Type 1 with One or Two *SMN2* Copies

Delivering AVXS-101 by Intravenous Infusion

**Summary of Changes:** Protocol Version 7.0, Amendment 6, 25 Jun 2020

Investigational Product: AVXS-101


This protocol amendment was required in order to:

- address COVID-19 related impact on trial conduct
- apply consistent definitions of the primary endpoint and exploratory endpoints
- clarify the collection and central review of videos of efficacy parameters
- clarify the schedule of assessments for some efficacy and safety parameters
- address specific requests from Competent Authorities regarding Safety Reporting timelines and Hy's Law Criteria
- clarify and correct statistical analysis definitions
- make administrative changes

The following changes were made to the Protocol from Version 6.0 Amendment 5 dated 26 Nov 2019 to Version 7.0 Amendment 6 dated 25 Jun 2020.

#### **SUMMARY OF CHANGES:**

The section below describes the changes incorporated into this version of the protocol.

Protocol Version 7.0 Incorporating Amendment 6 includes the following changes:

| <b>Description of Change</b> | Location(s) | Rational for Change |
|---|---|---|
| Updated protocol version, amendment number and date | Cover page and header throughout | Updated document |
| Replaced Corrected/updated s job titles | Signature page | To update per company administrative changes |
| Updated study physician email address Replaced Serious Adverse Event Reporting email and fax number | Key contact information | Updated contact details Updated following migration to Novartis safety database and reporting process |
| Addition of ADL (activities of daily living) Addition of AT (aminotransferase) and TBL (total bilirubin) | Section 4: List of Abbreviations and Definitions of Terms | As referenced in Section 13.1.1 Adverse Event (Table 4) and Section 14.4.1 Hy's Law Criteria |
| Text added to allow changes in study conduct during the COVID-19 pandemic (or other similar catastrophic event): - change to the conduct of study visits - when a subject may be considered withdrawn due | Section 7.1: Overall Trial Design<br>Section 8.3: Patient Withdrawal<br>Criteria<br>Section 11: Assessment of Efficacy<br>Section 12: Assessment of Safety<br>Section 16.1: Trial Monitoring<br>Section 18.3: Written Informed<br>Consent | In order to address the impact of the COVID-19 pandemic (or other similar catastrophic event) on: - a site's ability to conduct on-site study visits and efficacy and safety assessments per protocol |

Investigational Product: AVXS-101

| scription of Change | | |
|---|---|---|
| these factors, versus | Location(s) | Rational for Change - a subject's willingness |
| withdrawn consent | | or ability to continue |
| change to the manner in | | participating in the study |
| which efficacy and safety | | - a monitor's ability to |
| assessments are performed | | perform on-site |
| change to the manner in | | monitoring visits |
| which monitoring visits are | | - a site's ability to follow |
| performed | | the usual process of |
| the process of obtaining | | obtaining written |
| remote informed consent | | informed consent |
| dition of 'developmental' | Throughout | For consistency and |
| | Throughout | For consistency and |
| | | clarification |
| | Synopsis: Objectives: Exploratory | To align with Appendix 4 |
| | | 10 angh with rippendix |
| | 1 0 | |
| | | Updated information |
| | Section 5.5: Risks | At the request of the |
| | Section 11.1: Developmental | For clarification |
| • | | |
| xt was added to define the | Section 11.2.1: World Health | For clarification and to avoid |
| | | confusion between WHO |
| HO milestones | Reference Milestones | |
| | | milestones |
| leo Manual changed to | Throughout | |
| | 5 | Manual is the new reference |
| ·· | | document for Clinical |
| xt was added to clarify the | Section 11.2.2: Bayley Scales for | For clarification |
| ess at every visit, including at | Milestones | |
| finition of sitting relopmental milestones: HO – sitting without support ID #26 – functional ependent sitting ret for exploratory ectives/endpoints was revised include BSIDv03 Gross retor Subset Items 33, 34, 37, 42 regard to the date of the most ent data cut-off for safety a review from 08 March regard to 31 December 2019 retion 14.4.1 Hy's Law teria and definition inserted, ha link in Section 5.5 ret was added to state that at the months of age visit all relopmental milestones reduced regardless of revious attainment ret was added to define the reria required to attain each HO milestones reduced Manual changed to residual changed to res | Synopsis: Objectives: Exploratory Synopsis: Endpoint: Exploratory Section 6.3: Exploratory Objectives Section 14.1.1.1.3: Exploratory Endpoints Section 5.5: Risks Section 5.5: Risks Section 14.4: Safety Analysis Section 11.1: Developmental Milestones Section 11.2.1: World Health Organization Multicentre Growth Reference Milestones Throughout Section 11.2.2: Bayley Scales for Infant and Toddler Development/Developmental | Clarification For consistency and clarification To align with Appendix 4 Updated information At the request of the Belgium FAMPH For clarification For clarification and to aveconfusion between WHO and BSIDv03 gross motor milestones The Physical Assessments Manual is the new reference |

Investigational Product: AVXS-101

| <b>Description of Change</b> | Location(s) | Rational for Change |
|---|---|---|
| Month 18 regardless of previous attainment. Text added to clarify that Bayley Scales will be video recorded and videos containing developmental milestone evidence will be submitted for central review | Godina 11 2 2 Postor Contra for | |
| Text regarding the requirement to video record the Bayley Scales was deleted as this information is captured in 11.1 and 11.3 | Section 11.2.2: Bayley Scales for Infant and Toddler Development/Developmental Milestones | For clarification |
| Text added to state that additional information on contractures will also be collected, as described in the Physical Assessments Manual | Section 11.2.3: CHOP-INTEND | Collection of contractures data was included in the scoring sheet provided in Appendix 6 of previous protocol versions, but is not included in the new scoring sheet provided by CHOP. The Physical Assessment Manual contains a supplemental CHOP-INTEND contractures data collection sheet for use by investigator sites, to ensure consistency in the data collected throughout the study |
| Removal of text stating that each CHOP-INTEND exam will be submitted for review by central reviewer | Section 11.2.3: CHOP-INTEND | It was never the intention for CHOP-INTEND videos to be centrally reviewed |
| Text added to clarify that all videos of Developmental Milestones which meet WHO and BSID criteria will be provided to an independent central reviewer | Section 11.3: Video Evidence | For clarification |
| Text added to clarify that at the 18 month of age visit, the WHO Motor Developmental Milestone for sitting without support for at least 10 seconds and the BSID GM #26 sitting milestones will be submitted for central review, even if previously confirmed. | Section 11.3: Video Evidence | Only the WHO sitting milestone (primary endpoint) and BSID GM #26 sitting milestone (exploratory endpoint), and new developmental milestones attained for the first time, will be centrally |

Investigational Product: AVXS-101

| <b>Description of Change</b> | Location(s) | Rational for Change |
|---|---|---|
| New developmental milestones<br>attained for the first time at 18<br>months of age will also be<br>submitted for central review | | reviewed at the 18 months of age visit |
| Changed the form provided from 'by the Contract Research Organization' to 'by AveXis' | Section 13.1.2: Serious Adverse<br>Event<br>Section 13.1.3: Adverse Events of<br>Special Interest | SAE forms are now provided by AveXis using the Novartis template |
| Text added to clarify the reporting timelines for fatal/life threatening SUSARs | Section 13.5: Expedited Safety<br>Reporting to Regulatory Authorities | Per France ANSM request<br>and EU reporting<br>requirements |
| Text 'and subgroup analyses' removed Text 'and summarized by subgroup and overall' removed | Section 14.1.1.2.1: Intent-to-Treat<br>Population<br>Section 14.4: Safety Analysis | There is no subgroup<br>defined in the protocol; this<br>will be defined in the<br>Statistical Analysis Plan |
| One-sided exact binomial tests alpha level changed from 0.05 to 0.025 | Section 14.3.2: Primary and<br>Secondary Efficacy Analysis | Correction made to be consistent with power calculation |
| Schedule of Assessments was updated with a new line to specify the schedule of BSIDv03 Gross and Fine Motor Subtests (with video) | Appendix 1: Schedule of Assessments | To align with Section 11.2.2 |
| Notes for 12-Lead ECG,<br>Echocardiogram and 24-hour<br>Holter Monitor – (X) to be<br>completed every 3 months,<br>starting at Month 3 <u>until 12</u><br>months post-dose. | Appendix 1: Schedule of Assessments | For clarification. Because of the age of some subjects when they are dosed, they may not have visits at Months 9 or 12. It is important that these tests are performed every 3 months from Month 3 until 12 months post-dose, regardless of the visit/month number |
| Addition of copyright information at the bottom of each page of the Bayley record | Appendix 3: Bayley Scales of Infant and Toddler Development (Version 3) | Per copyright requirements |
| Source reference in footer changed from (36) to (38) | Appendix 5: Performance Criteria<br>for World Health Organization<br>(WHO) Developmental Milestones | Correction |
| Scoring sheet has been replaced with an updated version | Appendix 6: CHOP-INTEND | A new scoring sheet was provided by CHOP |